## **Cover Page**

Protocol Title: A randomized controlled post-market study to assess the impact of

peripheral intravenous catheter length and gauge on catheter indwell duration and haemolysis in human participants using a bilateral, cephalic

vein cannulation model.

Document Type: Statistical Analysis Plan

Document Date: 17-Mar-2021

NCT number: NCT04344314

## Global Clinical Development

Template GCD-3300.T01 Revision 01



## Statistical Analysis Plan

| Protocol Number/Version | BDT-19PIVCAU001 |
|---|---|
| Protocol Title | A randomized controlled post-market study to assess the impact of periph- |
| | eral intravenous catheter length and gauge on catheter indwell duration and |
| | haemolysis in human participants using a bilateral, cephalic vein cannulation |
| | model. |
| SAP Date | 17 Mar 2021 |
| Current Version | Version 1.0 |
| Version History | |

This document is proprietary to Becton Dickinson. No part of it may be distributed or shared with persons other than BD associates without written permission from Global Clinical Development (GCD).



## Approval

| Individual or Function | Name | Signature/Date |
|---|---|---|
| Statistician (Author) | Didier Morel | This document is signed electronically in the |
| | | eTMF system |
| R&D Study Lead | Christopher Rini | This document is signed electronically in the |
| | | eTMF system |
| Medical Affairs Team | Vincenzo Mancini | |
| Representative | | |
| Project Manager | Erin White | This document is signed electronically in the |
| | | eTMF system |
| Statistics Functional Manager | Ying Wan | This document is signed electronically in the |
| | | eTMF system |



## Contents

| 1.2 Objectives 1.2.1 Primary Objectives 1.2.2 Secondary Objectives 1.2.3 Exploratory Objectives 1.2.3 Exploratory Objectives 1.2.3 Exploratory Objectives 2.2 Study Description 2.1 Study Design 2.2 Study Population 2.2.1 Inclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.3.2 Blinding/Masking 1 2.3.2 Blinding/Masking 1 2.3.2 Blinding/Masking 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.5 Interim Analysis 1 2.5 Interim Analysis 1 2.5 Interim Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8 3 Exploratory Endpoints 1 2.5 Acceptance Criteria 1 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4 1 1 1 1 1 1 1 1 | 1 | $\operatorname{Intr}$ | roduction |
|---|---|---|---|
| 1.2.1 Primary Objectives 1.2.2 Secondary Objectives 1.2.3 Exploratory Objectives 1.2.3 Exploratory Objectives 2 Study Description 2.1 Study Design 2.2 Study Population 2.2.1 Inclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.3.3 Randomization and Blinding 1 2.3.1 Randomization 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.3.3 Procedures for Unblinding 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.5 Interim Analysis 1 2.5 Interim Analysis 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.1 Primary Endpoints 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.1 Endpoints 1 2.8.1 Endpoints 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.4 Exploration Definitions 1 2.8.4 Exploration Definitions 1 2.8.4 Exploration Definitions 1 2.8.4 Exploration Definitions 1 2.8.4 Exploration Definitions 1 2.8.4 Explorations 1 2.8.4 Exploration Definitions 1 2.8.4 Explorations 2 2 2 2 2 2 2 2 2 | | 1.1 | Background and Rationale |
| 1.2.2 Secondary Objectives 1.2.3 Exploratory Objectives | | 1.2 | Objectives |
| 1.2.3 Exploratory Objectives | | | 1.2.1 Primary Objectives |
| Study Description 2.1 Study Design 2.2 Study Population 2.2.1 Inclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.3.1 Randomization and Blinding 1 2.3.1 Randomization 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.6 Preliminary Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.1 Primary Endpoints 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 2.8.3 Exploratory Endpoints 2.8.3 Exploratory Endpoints 2.8.3 Exp | | | 1.2.2 Secondary Objectives |
| 2.1 Study Design 1 2.2 Study Population 1 2.2.1 Inclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.3 Randomization and Blinding 1 2.3.1 Randomization 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 | | | 1.2.3 Exploratory Objectives |
| 2.1 Study Design 1 2.2 Study Population 1 2.2.1 Inclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.3 Randomization and Blinding 1 2.3.1 Randomization 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 | | | |
| 2.2.1 Inclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.3 Randomization and Blinding 1 2.3.1 Randomization 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.1 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.7 Flush pressure profile and duration of flush 1 5.2.1 Sta | 2 | | |
| 2.2.1 Inclusion Criteria 1 2.2.2 Exclusion Criteria 1 2.3 Randomization and Blinding 1 2.3.1 Randomization 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio | | | · |
| 2.2.2 Exclusion Criteria 1 2.3 Randomization and Blinding 1 2.3.1 Randomization 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2.1 Stat | | 2.2 | · · |
| 2.3 Randomization and Blinding 1 2.3.1 Randomization 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1.1 Indwel | | | |
| 2.3.1 Randomization 1 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1. Indwell Time 1 5.2.1.2 Additional Descri | | | |
| 2.3.2 Blinding/Masking 1 2.3.3 Procedures for Unblinding 1 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flo | | 2.3 | Randomization and Blinding |
| 2.3.3 Procedures for Unblinding 1 | | | 2.3.1 Randomization |
| 2.4 Sample Size 1 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.2 Dominant arm 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2.1 | | | 2.3.2 Blinding/Masking |
| 2.5 Interim Analysis 1 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | 2.3.3 Procedures for Unblinding |
| 2.6 Preliminary Analysis 1 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 </td <td></td> <td>2.4</td> <td>Sample Size</td> | | 2.4 | Sample Size |
| 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | 2.5 | Interim Analysis |
| 2.7 Study Procedure 1 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | 2.6 | Preliminary Analysis |
| 2.8 Endpoints 1 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes | | 2.7 | · · |
| 2.8.1 Primary Endpoint 1 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | 2.8 | v |
| 2.8.2 Secondary Endpoints 1 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1. Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | • |
| 2.8.3 Exploratory Endpoints 1 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | |
| 2.9 Acceptance Criteria 1 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | |
| 3 Intended Statistical Software and Data Information 1 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | 2.9 | |
| 4 Analysis Population Set(s) 1 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | 12000p0a1200 011021a |
| 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | 3 | Inte | ended Statistical Software and Data Information |
| 4.1 Population Definitions 1 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | 4 | Ana | alysis Population Set(s) |
| 5 Statistical Analysis/Calculations 1 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | |
| 5.1 Derived Variables 1 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | • |
| 5.1.1 Haemolysis: Quantification and frequency of occurrence 1 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | 5 | Stat | |
| 5.1.2 Dominant arm 1 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | 5.1 | Derived Variables |
| 5.1.3 Blood draw fill time 1 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | 5.1.1 Haemolysis: Quantification and frequency of occurrence |
| 5.1.4 Intravenous thrombus 1 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | 5.1.2 Dominant arm |
| 5.1.5 Vessel diameter, Catheter to vein ratio 1 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | 5.1.3 Blood draw fill time |
| 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | 5.1.4 Intravenous thrombus |
| 5.1.6 Blood flow velocity 1 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | 5.1.5 Vessel diameter, Catheter to vein ratio |
| 5.1.7 Flush pressure profile and duration of flush 1 5.2 Analysis Methods 1 5.2.1 Statistical Analysis of Primary Endpoint 1 5.2.1.1 Indwell Time 1 5.2.1.2 Additional Description of Failure Modes 1 | | | , and the second se |
| 5.2 Analysis Methods | | | v |
| 5.2.1 Statistical Analysis of Primary Endpoint | | 5.2 | |
| 5.2.1.1 Indwell Time | | J. <u>-</u> | |
| 5.2.1.2 Additional Description of Failure Modes | | | v - |
| <u>.</u> | | | |
| | | | 1 |



| | | 5.2.2 | | al Analysis of Secondary Endpoints | 17 |
|---|---|---|---|---|---|
| | | | 5.2.2.1 | Haemolysis | 17 |
| | | | 5.2.2.2 | Blood draw fill time | 19 |
| | | | 5.2.2.3 | Relationship between catheter blood draw patency indwell time and pres- | |
| | | | | ence of intra/extravenous thrombi, thrombus length, thrombus type catheter | r |
| | | | | angle/tip location in situ, catheter length in vessel, vein depth from skin | |
| | | | | surface, C/V ratio, and vessel anatomy | 19 |
| | | | 5.2.2.4 | Evaluation of changes in vessel dimensions, PIVC position (insertion angle | |
| | | | | and in situ tip position), and haemodynamics from baseline throughout | |
| | | | | indwell time | 20 |
| | | 5.2.3 | Statistic | al Analysis of Exploratory Endpoints | 21 |
| | | 0.2.0 | 5.2.3.1 | Incidence of complications prompting device removal | 21 |
| | | | 5.2.3.2 | Flush pressure profile | 22 |
| | | 5.2.4 | | Considerations | $\frac{22}{22}$ |
| | | 5.2.4 $5.2.5$ | | hes and Analyses for Missing Data and Other Data Issues | 23 |
| | | 0.4.0 | Арргоас | nes and Analyses for Missing Data and Other Data Issues | 20 |
| 6 | Sum | mary o | f General | Study Data | 24 |
| | 6.1 | | | tion | 24 |
| | 6.2 | U | | ions | 25 |
| | | 6.2.1 | | eviations | 25 |
| | | 6.2.2 | | eviations | 25 |
| | 6.3 | Demos | | and Baseline Variables | 25 |
| | 6.4 | | | esses and Medical Conditions | 26 |
| | 6.5 | | | urrent Medications | 27 |
| | 6.6 | | | Malfunctions and Defects | 30 |
| | | | _ = =================================== | | |
| 7 | Safe | ty Anal | ysis | | 30 |
| _ | <b>.</b> . | | 1 · D1 | | |
| 8 | Inte | rim Ana | alysis Pla | $\mathbf{n}$ | 30 |
| 9 | Refe | rences | | | 31 |
| 10 | SAP | Revisi | on Histor | y | 32 |
| 11 | App | endix | | | 33 |
| <b>A</b> | Tabl | 0.0 | | | 33 |
| A. | | | rranhica | | 33 |
| | A.1<br>A.2 | _ | | History | 33 |
| | A.3 | · | | eteristics | 34 |
| | | | | Mode | $\frac{36}{37}$ |
| | A.5 | | | Mode | |
| | A.6 | | | Mode Per Day | 38 |
| | A.7 | | | ation | 40 |
| | A.8 | | | | 41 |
| | A.9 | | Draw Fil | l Time | 44 |
| | | | 1110 I 1001 | (TTT()T)(A() | /11 |



| $\mathbf{B}$ | Figu | res | 50 |
|--------------|-------|------------------------------------------|----|
| | B.1 | Survival | 50 |
| | B.2 | Indwell Time | 51 |
| | B.3 | Blood Analysis | 52 |
| | | B.3.1 cfHb | 52 |
| | B.4 | Haemolysis Occurrence | 54 |
| | B.5 | Blood Draw Fill Time | 56 |
| | B.6 | Thrombus Occurrence | 30 |
| | B.7 | Feature Importance with Boruta Algorithm | 32 |
| $\mathbf{C}$ | Listi | ings | 64 |
| D | Add | itional Figures | 72 |
| | D.1 | PIVC Rescue Decision Tree | 72 |



# List of Figures

| | 2.4.1 Details of sample size calculation | 11 |
|---|---|---|
| | 6.1.1 Skeleton flow diagram depicting participant disposition | 24 |
| | B.1.1Survival Curve for Indwell Time per Device Configuration | 50 |
| | B.2.1Boxplot for Indwell Time per Device Configuration | 51 |
| | B.3.1Boxplot for cfHb per Device Configuration for each Timepoint | 52 |
| | B.3.2Lineplot for cfHb per subject and Device Configuration over time | 53 |
| | B.4.1Barplot for Haemolysis Occurence (assessed with AU480) per Device Configuration B.4.2Barplot for Haemolysis Occurence (AU480 measurements) per Device Configuration for | 54 |
| | each Timepoint | 55 |
| | B.5.1Boxplot for Blood Draw Fill Time per Device Configuration | 56 |
| | B.5.2Estimated Blood Draw Fill Time Difference between Device Configurations for 2 and 6mL Vacutainer tubes | 57 |
| | B.5.3Lineplot for Blood Draw Fill Time per Device Configuration at each captured timepoint . B.5.4Estimated Blood Draw Fill Time Difference between Device Configurations for 2 and 6mL | 58 |
| | Vacutainer tubes per Time Point | 59 |
| | B.6.1Barplot for Thrombus Occurence per Device Configuration | 60 |
| | B.6.2Barplot for Thrombus Occurence per Device Configuration for each Timepoint | 61 |
| | B.7.1Boruta plot showing survival predictive importance of features | 62 |
| | B.7.2Boruta plot showing evolution of predictive importance of features over time | 63 |
| | D.1.1PIVC Rescue Decision Tree for Flush Procedures | 72 |
| | D.1.2PIVC Rescue Decision Tree for Aspiration Procedures | 73 |
| _ | | 10 |
| L | ist of Tables | |
| | 2.7.1 List of sampling time points for primary, secondary, and exploratory endpoints | 13 |
| | 6.4.1 List of medical conditions that will exclude participants from participating in this trial | 26 |
| | 6.5.1 List of current drug use resulting in exclusion $(1/2)$ | 27 |
| | 6.5.2 List of current drug use resulting in exclusion $(2/2)$ | 29 |
| | 6.5.3 List of current drug use trigerring deeper investigation for their effect on platelet function/thrombosis | 30 |
| | A.1.1Numerical Summary of Subjects Demographics, per Group (i.e. Gauge) and Overall | 33 |
| | A.2.1Numerical Summary of Familiy Medical History, per Group (i.e. Gauge) and Overall | 33 |
| | A.2.1Numerical Summary of Family Medical History, per Group (i.e. Gauge) and Overall | 00 |
| | continued | 34 |
| | A.3.1Numerical Summary of Baseline PIVC Characteristics, per Group (i.e. Gauge) and Overall | |
| | A.3.2Numerical Summary of Baseline Venipuncture Blood Analysis, per Group (i.e. Gauge) and | 94 |
| | Overall | 34 |
| | A.3.2Numerical Summary of Baseline Venipuncture Blood Analysis, per Group (i.e. Gauge) and | 34 |
| | Overall continued | 25 |
| | A.4.1Numerical Summary of Subjects Indwell Time in hours, per Device Configuration (Gauge | 35 |
| | and Length) and Overall | 36 |
| | A.4.2Proportional Hazard Ratios computed from Cox Proportional Hazards model for Indwell | |
| | time | 36 |
| | A.5.1Failure Modes Count Overall | 37 |
| | A.5.2Failure Modes Count Per Device Configuration | 37 |
| | A.6.1Failure Modes Count Overall Per Day | 38 |



| A.6.2Failure Modes Count Per Device Configuration | 39 |
|---|---|
| A.7.1Remediation Steps Count Overall | 40 |
| A.7.2Remediation Characteristics Count per Device Configuration per Day | 40 |
| A.8.1Numerical Summary of Subjects Blood Analysis, for each time point, per Device Configu- | |
| ration (Gauge and Length) and Vacutainer tube and Overall | 41 |
| A.8.1Numerical Summary of Subjects Blood Analysis, for each time point, per Device Configu- | |
| ration (Gauge and Length) and Vacutainer tube and Overall continued | 42 |
| A.8.1Numerical Summary of Subjects Blood Analysis, for each time point, per Device Configu- | |
| ration (Gauge and Length) and Vacutainer tube and Overall continued | 43 |
| A.9.1Numerical Summary of Blood Draw Fill Time in seconds for each Vacutainer tube, per | |
| Device Configuration (Gauge and Length) and Overall | 44 |
| A.9.2Numerical Summary of Blood Draw Fill Time in seconds for each Vacutainer tube, for | |
| each time point, per Device Configuration (Gauge and Length) and Vacutainer tube and | |
| Overall | 44 |
| A.9.2Numerical Summary of Blood Draw Fill Time in seconds for each Vacutainer tube, for | |
| each time point, per Device Configuration (Gauge and Length) and Vacutainer tube and | |
| | 45 |
| A.9.2Numerical Summary of Blood Draw Fill Time in seconds for each Vacutainer tube, for | |
| each time point, per Device Configuration (Gauge and Length) and Vacutainer tube and | |
| Overall continued | 46 |
| A.9.3ANOVA table for Blood Draw Duration linear mixed effect model | 47 |
| A.9.4Multiple Comparisons Based on linear mixed effect model for Blood Draw Duration. | |
| Sidak's adjustement for multiple comparisons was used | 47 |
| A.10. Numerical Summary of Thrombus Occurrence, per Device Configuration (Gauge and Length) | |
| and Overall | 49 |
| A.10. Numerical Summary of Thrombus Analysis, for each time point, per Device Configuration | |
| (Gauge and Length) and Overall | 49 |
| C.0.1Dummy randomization list (rows 1 to 40) | 64 |
| C.0.2Dummy Demographics listing (rows 1 to 40) | 65 |
| C.0.3Dummy Family Medical History listing (rows 1 to 40) | 66 |
| C.0.4Dummy Baseline listing (rows 1 to 40) | 67 |
| C.0.5Dummy Indwell Time listing (rows 1 to 40) | 68 |
| C.0.6Dummy Blood Analysis listing (rows 1 to 40) | 69 |
| C.0.7Dummy Blood Analysis Baseline listing (rows 1 to 40) | 70 |



## List of Abbreviations and Definitions

- BD: Becton Dickinson and Company
- BMI: Body Mass Index
- cfHb: Cell-free hemoglobin
- CI: Confidence Interval
- CRF: Case Report/Record Form
- CTU: Clinical Trials Unit
- C/V: Catheter to vein ratio
- Device Configuration: One of the following combinations of gauge and length
  - 22G & 1 inch
  - 22G & 1.75 inch
  - 20G & 1 inch
  - 20G & 1.75 inch
- eCRF: Electronic Case Report/Record Form
- FDAAA: FDA Amendments Act of 2007
- GCP: Good Clinical Practice
- GCUH: Gold Coast University Hospital
- HIV: Human Immunodeficiency Virus
- IRB/HREC: Institutional Review Board/Human Research Ethics Committee
- LLAD: Luer Lok Access Device
- PIVC: Peripheral intravenous catheter
- **PWD:** Pulse Wave Doppler
- SD: Standard Deviation
- **SOP:** Standard Operating Procedure
- XLabS: Experimental laboratory science group



## 1 Introduction

#### 1.1 Background and Rationale

BD is investigating a specific PIVC device design factor (length and gauge) that may extend indwell time and consequently enable successful PIVC use (i.e. blood collection) throughout dwell time. Identifying device design factors that increase PIVC dwell time and reduce incidence of haemolysis would reduce associated workload costs (e.g., recollection of hemoglobin-free serum samples, PIVC reinsertion) for healthcare institutions.

#### 1.2 Objectives

#### 1.2.1 Primary Objectives

To assess patent indwell time for PIVCs of different length and gauge.

#### 1.2.2 Secondary Objectives

- To assess haemolysis occurrence based on blood collection device, catheter device configuration.
- To evaluate blood draw fill time
- To determine the relationship, if any, between catheter blood draw patency indwell time and presence of intra/extravenous thrombi, catheter angle/tip location in situ, catheter length in vessel, vein depth from skin surface, C/V ratio, and vessel anatomy
- To evaluate changes in vessel dimensions, PIVC position (insertion angle and *in situ* tip position), and hemodynamics from baseline throughout indwell time

## 1.2.3 Exploratory Objectives

- To assess incidence of complications prompting device removal
- To evaluate manual flush variability (as applicable) using in-line pressure measurements

## 2 Study Description

#### 2.1 Study Design

This is a single-center, open-label, multi-visit, self-controlled study design, in 40 healthy participants, randomized by gauge of peripheral intravenous catheter (PIVC) device into the lower arm cephalic vein of both arms. The purpose of this feasibility study is to assess impact of catheter length and gauge on PIVC indwell time over a multi-day (72 hour) period. This study will also evaluate the incidence of haemolysis from PIVC using a LLAD and vacutainer tube (2mL, 6mL) blood collection method compared to venipuncture from the antecubital fossa.

#### 2.2 Study Population

Participants of clinical trials at the Clinical Trials Unit (CTU) based at the Griffith University Gold Coast campus are recruited through two primary mechanisms: 1) local advertising via digital and paper flyers; and 2) identification of suitable participants in the CTU volunteer registry (database). All advertising in the printed and audio-visual media has prior approval of the Griffith University Human Research Ethics Committee (HREC). The CTU volunteer registry has been maintained since 2015 and currently contains more than 700 volunteers.

Participants not meeting all criteria will be assessed by a medical monitor and included if patient safety is not adversely impacted.



#### 2.2.1 Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

- Female or Male
- 18-65 years of age
- Not pregnant at time of recruitment within 48 hrs Day 1 procedures (self-reported)
- Normal coagulation results (prothrombin time 13-17 sec; activated partial thromboplastin time 27-37 sec)
- Normal platelet aggregation results for ADP, TRAP, and collagen induced maximal amplitude (>70% amplitude over 6 mins)
- Target cephalic veins readily cannulatable (i.e.,  $\geq \sim 2.55$  mm to obtain C/V ratio less than 45% as indicated by standard 52 of the INS guidelines
- Able and willing to provide verbal and written consent
- Current Medicare card holder

#### 2.2.2 Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

- History of pro coagulative state/condition (e.g. previous deep vein thrombosis)
- Current hypertension (e.g., systolic >139 OR diastolic >89 mmHg)
- Currently on any anti-coagulant or platelet inhibitor medication. Use of NSAIDs and aspirin will be documented however not exclusionary.
- Hemophilia or any current or history of bleeding disorder or tendency
- Presence or report of current blood borne disease/infection (e.g. hepatitis, HIV, leukemia, lymphoma)
- Difficult vascular access (i.e., vein must be readily palpable and cannulatable no less than  $\sim 2.55$  mm diameter to maintain  $\leq 45\%$  C/V ratio) as indicated by standard 52 of the INS guidelines 27
- Allergy or sensitivity to chlorhexidine gluconate, isopropyl alcohol, latex, or skin adhesives
- BMI  $<18.5 \text{ kg/m}^2 \text{ or } >35 \text{ kg/m}^2$
- Positive results for the urine drug screen at screening or check-in (including opiates, methadone, cocaine, amphetamines)
- History or presence of alcoholism (self-reported) or drug abuse within the past 2 years
- A current or previous medical, physical, mental/cognitive disorders or anatomical conditions that, in the opinion of the investigator, would place the patient at risk, would make them unable to perform study procedures or has the potential to confound interpretation of the study results (e.g., musculo-skeletal injury, chronic back pain)
- Employed by Becton Dickinson, Teleflex Medical, Smiths Medical or B Braun (conflict of interest)

#### 2.3 Randomization and Blinding

#### 2.3.1 Randomization

Participants will be randomized using R statistical software (R 3.6.2 or higher). The generation of the randomization list will be conducted by a staff member not involved in data acquisition or analysis. Each randomization number will have a corresponding code (e.g., LA\_20G\_1.75 - indicating a Nexiva 20G 1.75 will be first inserted into the left arm). The participant will then have the other length PIVC of the same gauge inserted into the contralateral arm. Intervention kits will be created for each participant

using large ziplock bags with all necessary (plus extra) consumables inside. Each kit will be separated via separate ziplock bags into consumables required for the right arm and left arm. Once the kits have been created, the appropriate randomization number will be recorded on the outside of each. Subsequently,



the corresponding code will be placed in an envelope and sealed with the randomization number written on the outside of the envelope. These envelopes will be produced in duplicate with the second envelope sealed in a locked cabinet in the CTU for the circumstance where unblinding is required. Thereafter, the randomization list excluding the corresponding code will be given to the postdoctoral research fellow for storage until a randomization number is requested for the study.

#### 2.3.2 Blinding/Masking

Due to the concealment of intervention allocation, most staff members, other than the inserter and study manager (research assistant), will be blinded to which gauge and length catheter the participant is receiving. In order to avoid bias, sonographic data measurements (e.g., vessel diameter, C/V ratio, blood flow velocity) will be acquired on a separate day at the end of each working week. The acquisition of the sonographic measurements will be conducted by the sonographer). All concealed data will be transferred into an Excel spreadsheet that will be subsequently grouped into 2 groups in a separate Excel spreadsheet by a staff member not involved in data analysis and is unblinded. This will allow the researchers to analyze the data without having access to information about the allocation

#### 2.3.3 Procedures for Unblinding

In the unlikely scenario of a SAE, the study manager or post-doctoral research fellow will open the duplicate envelope located in the locked cabinet of the CTU that has the randomization number written on the outside and contains the corresponding code within. The information will be provided to any personnel that require the information (e.g., the study Medical Doctor) as deemed necessary by the Principal Investigator.

#### 2.4 Sample Size

There is limited published data investigating the impact of PIVC catheter length on indwell time; a single article was found in the literature comparing catheter survival between a BD PIVC catheter (20 gauge; 4.78 cm/1.88-inch length) and midline catheter (POWERWAND<sup>TM</sup>, 19.5 gauge; 6 cm/2.3-inch length). The indwell time results for this research were utilized to calculate a sample size estimate using the routine "Survival - Two Survival Curves - Logrank Tests" available in the software PASS 2019. Based on the available dataset, a sample size of  $\sim 20$  participants per PIVC length would be required, considering median failure times of catheter of different lengths of 1 and 3 days, as can be seen in Figure 2.4.1. The same calculation will be applied to investigating the impact of increased gauge, because the increased volume of catheters is similar in both condition (i.e., 1 versus 1.75 inch = 75% increased volume; 20 versus 22 gauge = 51% increased volume).

Figure 2.4.1: Details of sample size calculation

Logrank Tests Numeric Results for the Logrank Test in Terms of Sample Size Alternative Hypothesis: Two-Sided Ctrl Trt Acc-Med Med rual Ctrl Trt Haz Surv Surv Acc. Time Ctrl Ratio Time Time rual Total Trt to to (HR) (M2)Pat'n Loss Loss Trt Ctrl Alpha Power (M1)Time 0.8054 39 0.3333 1.00 3.00 Equal 0/3 0.0000 0.0000 0.0000 0.0000 0.0500 0.1946



#### 2.5 Interim Analysis

A formal interim analysis is not planned. However, after 5 participants have completed their follow-up visit (V6), the in-situ catheter positions will be compared to the expected position based on the catheter lengths. Only summary statistics related to the catheter length will be provided (mean, median, percentage) and no statistical test will be performed.

#### 2.6 Preliminary Analysis

In order to answer critically urgent business questions, a preliminary analysis will be performed by an independent statistician prior to the final database lock. This analysis will be limited to the analysis of the following specific endpoints:

- Indwell time (as described in section 5.2.1.1) and ranking of factor influencing indwell time (as described in section 5.2.2.3 by item 7)
- Haemolysis as a continuous measurement by device configuration and over time, including baseline venipuncture rate as relative comparator, as described in section 5.2.2.1 by item 1 (including the preliminary Boruta analysis)
- Rate of occurrence of Haemolysis by device configuration and over time, including baseline venipuncture rate as relative comparator, as described in section 5.2.2.1 by item 2 (including the preliminary Boruta analysis)
- Thrombus observation by device configuration over time, as described in section 5.2.2.3 by items 1, 2, 3, 4 and 7
- Incidence of failure modes for device removal, as described in section 5.2.1.2

The results of the preliminary analysis will be communicated by the independent statistician to Christopher Rini (Associate Director - Biomedical Engineering) who will be responsible for sharing them with Jeff O'Bryan (Director - Product Development Engineering), select MDS designees, and Ron Pettis (Director/Principal Scientist - Parenteral Research). Preliminary analysis will not be shared beyond those required for making time-critical business decisions on behalf of the MDS business unit.

Every GCD employee involved in the study execution, especially the lead study statistician, as well as all site employees involved in the study execution, will remain blinded to the results of this preliminary analysis until database lock.

It is understood by all parties that the results of this primary analysis will be subject to confirmation after database lock and fulfillment of all the processes related to data quality described in the Data Management Plan.

#### 2.7 Study Procedure

The time-windows for collection of the primary, secondary and exploratory endpoints are detailed in Table 2.7.1.

The primary endpoint data (catheter dwell time) and exploratory endpoint data (PIVC complications) will be collected over 7 time-windows (see text highlighted in orange on Table 2.7.1). The secondary endpoint data (cfHb, blood draw time) will be collected over 8 discrete timepoints (including baseline, see text highlighted in red on Table 2.7.1).

All other secondary endpoint data (e.g., blood flow velocity, vessel diameter), except incidence of extravenous thrombus (assessed once the catheter is removed), will be collected over 15 timepoints (see text



highlighted in blue and grey on Table 2.7.1). Please note that the cells that indicate 'Day' in Table 1 are indicating the interventional visit days and are not inclusive of the screening visit or follow-up visit.

The flush pressure profile exploratory endpoint data will be collected over 7 timepoints (see text highlighted in blue on Table 2.7.1).

Table 2.7.1: List of sampling time points for primary, secondary, and exploratory endpoints. cfHb: cell-free hemoglobin; TIP: catheter tip position; BFV: blood flow velocity; C/V: catheter to vein ratio; PRES: in vivo pressure; PIVC: peripheral intravenous catheter; FILL: blood draw fill time. Time T+00:00 is the time of insertion

| Day | Visit | Timepoint code | $\begin{array}{c} {\rm Approximate} \\ {\rm (hh:mm)} \end{array}$ | Time | Measurements taken |
|---|---|---|---|---|---|
| | Baseline | D1.1 | T-00:60 | | TIP, BFV, C/V via ultrasound (no indwelling catheter) |
| | | D1.2 | T-00:40 | | cfHb via venipuncture |
| Day 1 | Manaira | D1.3 | T+00:15 | | TIP, BFV, $\mathrm{C/V}$ via ultrasound, PRES via PIVC during flush |
| Day 1 | Morning | D1.4 | T+00:25 | | cfHb, FILL via PIVC |
| | | D1.5 | T+00:35 | | TIP, BFV, C/V via ultrasound |
| | A Channa an | D1.6 | T+06:00 | | TIP, BFV, $C/V$ via ultrasound, PRES via PIVC during flush |
| | Afternoon | D1.7 | T+06:15 | | cfHb, FILL via PIVC |
| | | D1.8 | T+06:25 | | TIP, BFV, C/V via ultrasound |
| | 34 . | D2.1 | T+24:00 | | TIP, BFV, C/V via ultrasound, PRES via PIVC during flush |
| | Morning | D2.2 | T+24:15 | | cfHb, FILL via PIVC |
| Day 2 | | D2.3 | T+24:25 | | TIP, BFV, C/V via ultrasound |
| | Afternoon | D2.4 | T+30:00 | | TIP, BFV, $C/V$ via ultrasound, PRES via PIVC during flush |
| | | D2.5 | T+30:15 | | cfHb, FILL via PIVC |
| | | D2.6 | T+30:25 | | TIP, BFV, C/V via ultrasound |
| | Morning | D3.1 | T+48:00 | | TIP, BFV, $\mathrm{C/V}$ via ultrasound, PRES via PIVC during flush |
| | | D3.2 | T+48:15 | | cfHb, FILL via PIVC |
| Day 3 | | D3.3 | T+48:25 | | TIP, BFV, C/V via ultrasound |
| | A Ct annua an | D3.4 | T+54:00 | | TIP, BFV, $C/V$ via ultrasound, PRES via PIVC during flush |
| | Afternoon | D3.5 | T+54:15 | | cfHb, FILL via PIVC |
| | | D3.6 | T+54:25 | | TIP, BFV, C/V via ultrasound |
| Doy 4 | Morning | D4.1 | T+72:00 | | TIP, BFV, $C/V$ via ultrasound, PRES via PIVC during flush |
| Day 4 | Morning | D4.2 | T+72:15 | | cfHb, FILL via PIVC |
| | - | D4.3 | T+72:25 | - | TIP, BFV, C/V via ultrasound |



## 2.8 Endpoints

#### 2.8.1 Primary Endpoint

The primary endpoint is the catheter indwell time, defined as the time from catheter insertion to time of catheter failure. It is measured in hours.

#### 2.8.2 Secondary Endpoints

- Haemolysis measured in three different ways with cfHb, AU480 and visual assessment: Quantification of cell free hemoglobin and frequency of samples exceeding a concentration of 50 mg/dL.
- Blood draw fill time. Defined as the duration from attachment of vacutainer to time when blood fills to pre-defined fill level. It is measured in seconds.
- Relationship, if any, between catheter blood draw patency indwell time and presence of intra/extravenous thrombi, catheter angle/tip location in situ, catheter length in vessel, vein depth from skin surface, C/V ratio, and vessel anatomy assessed via the incidence of:
  - Intravenous thrombus (mural, at tip)
  - Vein collapse
  - Presence and location of a valve relative to catheter tip
  - Side branches relative to catheter tip detected through ultrasound
- Evaluation of changes in vessel dimensions (Catheter to vein ratio), PIVC position (insertion angle and *in situ* tip position), and hemodynamics from baseline throughout indwell time evaluated using:
  - Vessel diameter or Catheter to vein ratio (C/V ratio)
  - Blood flow velocity
  - In situ tip position
  - Extravenous thrombus visually observed upon device removal within:
    - \* Catheter hub
    - \* Needleless connector
    - \* Extension tubing via visual observation

#### 2.8.3 Exploratory Endpoints

- Incidence of complications prompting device removal assessed by the frequency of occurrence of the following events:
  - Vein collapse
  - Phlebitis
  - Venous thrombosis
  - Dislodgement
  - Infiltration (called Extravasation in the protocol)
  - Accidental removal
- Manual flush variability will be evaluated using duration of flush and characteristics of Flush pressure profile (peak force) obtained on in-line pressure measurements

#### 2.9 Acceptance Criteria

No acceptance criteria have been established for this study.

#### 3 Intended Statistical Software and Data Information

The analysis will be conducted with R version 4.0.3 (2020-10-10) [1] or a more recent version. The extraction of the pressure profile and duration of flush characteristics will be performed by BDTI R&D



using LabView 2020 with the script PIVC linedraw, version 1.1.2. Results will be provided to the study statistician in a csy file.

## 4 Analysis Population Set(s)

#### 4.1 Population Definitions

In the unforeseen circumstance of a protocol deviation (e.g., 20G PIVC instead of 22G PIVC; blood was collected into 6mL vacutainer before 2mL for a specific participant), the data will be analyzed "as treated" - that is, data will be analyzed as the participant's actual received intervention. However, in the unforeseen circumstance of a protocol deviation whereby a participant receives the wrong intervention (e.g., two different gauge catheters; two 20G catheters of the same length), they will be treated as per protocol (PP) and thus their data will be excluded from the study because paired comparison of catheter length will not be possible.

## 5 Statistical Analysis/Calculations

#### 5.1 Derived Variables

Below is a list of variables that require calculation or transformation of data that will be used for derived outcomes. Any variables that are not listed below do not have derived outcomes.

#### 5.1.1 Haemolysis: Quantification and frequency of occurrence

To quantify cfHb, whole blood collected and anticoagulated with Ethylenediaminetetraacetic acid (EDTA), will be centrifuged at 1200 x g for 10 min. The top half of the supernatant will be added to 0.01% Na<sub>2</sub>CO<sub>3</sub> (1:6) and the absorbance of each sample will be measured at 380, 415 and 450 nm using a spectrophotometer (MultiSkan GO, Thermo Fisher Scientific; MA, USA). The cfHb will subsequently be calculated from these absorbances using the Harboe method 45, as described in Equation 1.

$$cfHb\left(\frac{mg}{dL}\right) = \left(\frac{167.2Abs_{415} - 83.6Abs_{450} - 83.6Abs_{380}}{10}\right) \times \frac{1}{dilution in Na_2CO_3} \tag{1}$$

Additionally, an automated biochemistry analyzer (AU480, Beckman Coulter, USA) will be employed for a clinical measurement of haemolysis and assessing the frequency of cfHb above a threshold of 50 mg/dL. The accuracy of the device is not sensitive to measurements below 50 mg/dL. Lastly, visual assessment of haemolysis will be checked, and photographs taken of each sample.

#### 5.1.2 Dominant arm

The identification of the dominant will be performed for each subject crossing information from the VENIPUNCTURE CRF questions "Arm Venipuncture Performed from?" and "Was this the Non-Dominant Arm?", available in the variables DELOC and DENDARM, respectively, from the table VPVP.

#### 5.1.3 Blood draw fill time

The blood draw fill time (seconds) will be calculated manually using a stopwatch - from connection to blood reaching predetermined fill line.

#### 5.1.4 Intravenous thrombus

The presence of an intravenous thrombus (mural, at tip) will be ascertained using ultrasound.

#### 5.1.5 Vessel diameter, Catheter to vein ratio

The vessel diameter, and C/V ratio (Catheter to vein ratio) will be derived from the mean average of three cross-sectional, B-mode scans to be taken with the indwelling PIVC in view. The vessel diameter



will be calculated from the horizontal axis using the internal calculations of the ultrasound. The data will be reported as the average of the values taken from three images. The catheter diameter will be derived from the device specifications, where catheter outer diameter is reported to be 0.90 mm and 1.10 mm, respectively for 22G and 20G catheters.

#### 5.1.6 Blood flow velocity

The blood flow velocity calculations (i.e. maximum and mean velocity of 5 seconds of data) will be derived from the area underneath the velocity spectrum boundary using the internal measurement tool of the ultrasound.

#### 5.1.7 Flush pressure profile and duration of flush

The flush pressure profile (i.e. duration and peak pressure) will be derived from the pressure trace from a 3 to 10 mL saline flush performed upon first accessing the device at each time point indicated in Table 2.7.1. Pressure (P) will be recorded prior to commencement of the flush and this will be defined as "baseline" pressure. Commencement of the flush will induce a spike in positive pressure, and this will be defined as "time point zero"  $(t_0)$ . The time point at which the spike in positive pressure returns to baseline will indicate completion of the flush and will be defined as the "completion time point"  $(t_c)$ . Subsequently, the duration of the flush will be derived by subtracting time point zero from the completion time point, as described in Equation 2.

$$flush duration = t_c - t_0 (2)$$

Alternatively, the duration of the flush could be reduced to the time between the max pressure and the completion time point, as described in Equation 3.

alternative flush duration = 
$$t_{max} - t_0$$
 (3)

The pressure reading with the maximal value between the two time points will be recorded as the peak pressure, defined as in Equation 4.

flush peak pressure = 
$$\max_{t_0 < t < t_c} P(t)$$
 (4)

#### 5.2 Analysis Methods

The following section defines hypothesis that will be tested. However, given the feasibility nature of the study no acceptance criteria were defined and estimating absolute effects and statistical significance of difference between device configuration is of similar importance.

#### 5.2.1 Statistical Analysis of Primary Endpoint

#### **5.2.1.1** Indwell Time

It is hypothesized that:

- PIVC indwell time will be greater for longer catheters
- PIVC indwell time will be greater for catheters of smaller gauge (larger bore)

In order to test these hypotheses, catheter indwell time will be assessed using survival analysis, including:

- Kaplan-Meier survival curves including Log-Rank test p-value
- Cox Proportional Hazards Model with Hazard Ratios for each device vs. default device condition (BD Nexiva 20G x 1 inch) and associated 95% Confidence Intervals. Effect of the following covariates will be investigated: gender, age, BMI and dominant arm.



Main analysis will be performed stratified by device, depending on the results pooled analyses by gauge or by catheter length might be performed. An example of the Kaplan-Meier curve and associated metrics is provided in Appendix B by Figure B.1.1. An example of the Hazard Ratios extracted from the Cox Proportional Hazards models is provided in Appendix A by Table A.4.2.

For the purpose of this survival analysis, device failure (inability to flush or draw blood, see section 6.6) will be identified as follows:

- Blood Draw: Variables DEBLDCS equal to "N" and DEBLDRS equal to "N" from table INBCINBC
- Flush: Variables DEFLSSU equal to "N" and DEFLSRS equal to "N" from table INFL

Failure can occur during any of the 7 repeats of the blood draw (for either tube volumes) or flush processes, as highlighted in orange on Table 2.7.1, for right or left arm, per randomization schedule. Date-time of failure is then given by the aggregation of variables DEDTN & DEFTM, from tables INBCINBC or INFL, respectively for blood draw or flush.

Additional Indwell Time summary statistics and graphical representation will be provided as represented in Appendix A by Table A.4.1 and in Appendix B by Figure B.2.1, respectively.

#### 5.2.1.2 Additional Description of Failure Modes

Failure mode counts will be summarized overall, per device, per day and per device per day, as represented in Appendix A by Tables A.5.1, A.5.2, A.6.1 and A.6.2, respectively. A list of the failure modes available in the free form text field describing the "Other" category will be provided. Companion bar plots will be generated for each of these tables.

**Note:** It is possible that despite a failure having been observed during a 2mL, a draw was attempted at 6mL, such situation would result in failures being counted twice. To avoid this, any failure information with a time stamp ulterior to the time stamp associated with the first failure record will be discarded from the data used to generate the principal tables summarizing the count of failure modes. A separate table will included providing counts of consecutive failures (defined as a failure occurring in a 6mL draw when a failure has already been observed for the immediately preceding 2mL).

#### 5.2.1.3 Additional Description of Failure Remediation

Failure remediation counts, which steps are described in the PIVC rescue decision trees for flush and aspiration procedures represented in Appendix D by Figures D.1.1 and D.1.2, will be summarized for each step overall and per device per day, as represented in Appendix A by Tables A.7.1 and A.7.2, respectively.

## 5.2.2 Statistical Analysis of Secondary Endpoints

#### 5.2.2.1 Haemolysis

It is hypothesized that:

• The cfHb concentrations observed in blood samples (all vacutainers, at all timepoints) collected from shorter catheters will be greater than that observed in longer catheters.



- The cfHb observed in blood samples (all vacutainers, at all timepoints) collected from catheters with a larger gauge (smaller bore) will be greater than blood collected from smaller gauge (greater bore).
- The cfHb observed in blood samples (all catheters) collected into greater volume vacutainers will be greater than blood collected into smaller volume vacutainers.

#### Haemolysis will be assessed through:

- 1. Quantification of average cfHb concentrations measured at each time point listed in red in Table 2.7.1. A linear mixed effect model will be used with cfHb as response and subject as random effect. Time, gauge, length, vacutainer volume and baseline (at D1.2) cfHb (2ml, 6ml measures will be used as separate continuous variables and will be retained in the model if significant) will be fixed effects. An example of the summary statistics table and associated graphical representation are provided in Appendix A by Table A.10.2 and in Appendix B by Figure B.3.1, respectively.
- 2. Rate of occurrence measured using the results of the cfHb concentrations at each time point listed in red in Table 2.7.1. Samples will be considered positive for haemolysis for cfHb concentration ≥ 50mg/dL¹. A logistic mixed effect model will be used with haemolysis occurrence as response and subject as random effect. Time, gauge, length, vacutainer volume and baseline (at D1.2) cfHb will be fixed effects. Tables summarizing occurrence rates per device per time point and associated graphical representation will be similar to the one provided for rate of occurrence measured using the results of the AU480 analysis (see next item) in Appendix A by Table A.10.2 and in Appendix B by Figures B.4.1 and B.4.2, respectively. Contrast based multiple comparisons will be used to compare haemolysis rate between conditions (between gauge, between length) at each timepoint.
- 3. Rate of occurrence measured using the results of the AU480 Analysis at each time point listed in red in Table 2.7.1. Samples will be considered positive for haemolysis for AU480 output of + (50-99mg/dL), ++ (100-199mg/dL), +++ (200-299mg/dL), ++++ (300-500mg/dL) and +++++ (>500mg/dL), i.e. anything different from N (<50mg/dL)<sup>2</sup>. A logistic mixed effect model will be used with haemolysis occurrence as response and subject as random effect. Time, gauge, length, vacutainer volume and baseline (at D1.2) cfHb will be fixed effects. Examples of the table summarizing occurrence rates per device per time point and associated graphical representation are provided in Appendix A by Table A.10.2 and in Appendix B by Figures B.4.1 and B.4.2, respectively. Contrast based multiple comparisons will be used to compare haemolysis rate between conditions (between gauge, between length) at each timepoint.
- 4. Rate of occurrence measured using the results of the visual assessment at each time point listed in red in Table 2.7.1. Samples will be considered positive for haemolysis for visual values ≥ 50mg/dL, as shown on the reference chart. A logistic mixed effect model will be used with visually observed haemolysis occurrence as response and subject as random effect. Time, gauge, length, Vacutainer tube volume and baseline (at D1.2) cfHb will be fixed effects. An example of the table summarizing occurrence rates per device per time point is provided in Appendix A by Table A.10.2. Graphical representation will be similar to the ones given as example for the AU480 analysis. Contrast based multiple comparisons will be used to compare haemolysis rate between conditions (between gauge, between length) at each timepoint.

In each case, i.e. for cfHb, AU480 and visual assessment, modeling will be preceded by an assessment of the importance of potential covariates using the Boruta algorithm. The covariates of interest will include,

<sup>&</sup>lt;sup>1</sup>A separate assessment of the relationship between the cfHb and AU480 measurements will be performed in order to check the validity of this threshold, which could be modified upon review of these results.

<sup>&</sup>lt;sup>2</sup>A separate assessment of the relationship between the cfHb and AU480 measurements will be performed in order to check the validity of this threshold, which could be modified upon review of these results.



but will not be limited to:

- Presence of thrombus
- Size of thrombus
- Proximity of thrombus to tip of catheter
- Draw rate
- Screening Blood Testing (as provided by Blood Testing CRF)
  - Coagulation Panel: PT & aPTT
  - Platelet Aggregometry: ADP, TRAP & Collagen Induced Maximal Amplitude
  - Blood Screening: Blood Glucose & Triglycerides
  - Liver Panel: ALT Average Measurement & AST Average Measurement

The significance of the most important features will be assessed by inclusion in the corresponding models and only significant covariates will be retained in the final model.

#### 5.2.2.2 Blood draw fill time

It is hypothesized that:

- The blood draw duration observed for blood samples (all vacutainers, at all timepoints) collected from shorter catheters will be decreased when compared to longer catheters of the same gauge.
- The blood draw duration observed for blood samples (all vacutainers, at all timepoints) collected from smaller gauge (larger bore) catheters will be decreased when compared to larger gauge (smaller bore) catheters of the same length, over time.
- The blood draw duration observed for blood samples (all catheters, at all timepoints) collected into greater volume vacutainers will be increased when compared to smaller volume vacutainers.

A linear mixed effect model will be used with blood draw fill time as response and subject as random effect. Time, device configuration (gauge, length and their interaction), Vacutainer tube volume and baseline (at D1.2) blood draw fill time will be fixed effects. Contrast based multiple comparisons will be used to compare blood draw fill time between conditions (between gauge, between length) at each timepoint. Example tables for summary statistics (overall and per time point for each Vacutainer tube volume are given in the Appendix section by Table A.9.1 and Table A.9.2, respectively. Graphical representations of distribution of blood draw time per device is provided in Figure B.5.1 and of average blood draw time is shown in the Appendix section by Figure B.5.3. Example tables for ANOVA tables (Table A.9.3) and multiple comparisons (Table A.9.4) can be found in the Appendix A

# 5.2.2.3 Relationship between catheter blood draw patency indwell time and presence of intra/extravenous thrombi, thrombus length, thrombus type catheter angle/tip location *in situ*, catheter length in vessel, vein depth from skin surface, C/V ratio, and vessel anatomy

Relationship, if any, will be assessed through the computation of:

- 1. Summary statistics stratified by indwell time considered as a discrete variable (0, 6, 24, 30, 48, 54, 72 hours)
- 2. Scatter plot showing time between initial Thrombus observation to time of removal per Device Configuration
- 3. Bar plot showing percentage of thrombus for each time point per device configuration
- 4. Scatter plot showing thrombus length as a function of time grouped by device configuration
- 5. Relationship between flush technique and presence of Thrombus
- 6. Summary statistics and boxplot showing time between time of initial thrombus observation and device removal per device configuration



- 7. Importance of covariates will be computed with Boruta algorithm with a survival random forest model (an example output from the algorithm is provided in the Appendix by Figure B.7.1).
- 8. Test of predictive performance for the most important features (confirmed by the Boruta algorithm) using a leave-one-out strategy

In addition to the variables used in the primary endpoint survival model (device gauge and length), investigated baseline characteristics will be:

- Venous thrombosis
- Thrombus Length
- Thrombus Type
- Angles of insertion (Acute Inferior and Superior)
- Catheter to vein (C/V) ratio
- Catheter length in vessel
- Presence of side branches and/or intravenous valves
- Age
- Gender
- Height
- Weight
- BMI
- Dominant arm
- Medical history questionnaire responses
- Exploratory endpoints:
  - Vein collapse
  - Phlebitis
  - Dislodgement
  - Extravasation

item Screening Blood Testing (as provided by Blood Testing CRF)

- Coagulation Panel: PT & aPTT
- Platelet Aggregometry: ADP, TRAP & Collagen Induced Maximal Amplitude
- Blood Screening: Blood Glucose & Triglycerides
- Liver Panel: ALT Average Measurement & AST Average Measurement

The Boruta algorithm does not require specific formatting and generally works well with continuous and categorical variables. In some cases, it might be interesting to move from continuous format to a categorical one (e.g. age) depending on the final analysis. Categorization rules will be detailed whenever performed.

# 5.2.2.4 Evaluation of changes in vessel dimensions, PIVC position (insertion angle and *in situ* tip position), and haemodynamics from baseline throughout indwell time

These will be evaluated using:

- C/V ratio
- Catheter Length in Vessel (mm)
- Catheter Insertion Angle acute inferior border angle (deg)
- Catheter Insertion Angle acute superior border angle (deg)
- Blood Draw Time (sec)
- Blood Flow Velocity (cm/sec)
- In situ tip position (Mid-Stream & Wall Contact)



For each of these characteristics, summary statistics by indwell time considered as a discrete variable (0, 6, 24, 30, 48, 54, 72 hours) and line and bar plots will be generated on average for continuous and by proportion for categorical responses, respectively.

Line plots will be similar to the example provided for cfHb in Figure B.3.2 and bar plots will be similar to the example provided for Haemolysis occurrence in Figure B.4.1, both represented in Appendix B.

Mixed effect models will be used with corresponding response and subject as random effect. Time, gauge, length, Vacutainer tube volume and baseline measurement of response will be fixed effects. Depending on the type of the response variable, the models will be:

- Linear: C/V ratio, catheter length, catheter insertion angles and blood flow velocity
- Logistic: Tip positions

Depending on model results, contrast based multiple comparisons will be used to compare means between conditions (between gauge, between length) at each timepoint. Results will be provided in Tables similar to the example given for Blood Draw Fill time in Tables A.9.3 and A.9.4, as can be found in the Appendix A.

The relationship between C/V ratio and Blood Draw Time as well as between C/V ratio and Blood Flow Velocity will be investigate using relevant graphical representation (scatter plots) and measure of association.

#### 5.2.3 Statistical Analysis of Exploratory Endpoints

#### 5.2.3.1 Incidence of complications prompting device removal

Assessment of the incidence of reasons for removal, device handling descriptors and complication prompting device removal will include assessment of the frequency of occurrence of the following events:

- Reasons for removal:
  - End of study
  - Accidental Dislodgement
  - Flush Failure
  - Blood Draw Failure
  - Adverse Event
- Device handling descriptors:
  - Failure modes for Flush/Draw (2/6mL) by Device configuration
  - Success of specific remediation steps
  - Remediation occurrence rate by day and percentage of success
- Vein collapse
- Phlebitis
- Presence of Venous thrombosis
- Catheter Dislodgement from Vein
- Extravasation
- Accidental removal
- Catheter Dislodgement from Vein

For each of these characteristics, summary statistics by indwell time considered as a discrete variable (0, 6, 24, 30, 48, 54, 72 hours) and longitudinal line and bar plots will be generated on average for continuous and by proportion for categorical responses, respectively.



Lineplots will be similar to the example provided for cfHb in Figure B.3.2 and bar plots will be similar to the example provided for Haemolysis occurrence in Figure B.4.1, both represented in Appendix B.

Relationship between the occurrence of these events will be investigated using complementary approaches:

- Predictive Power over time (similar to Kramer's V but no need to transform variables)
- Boruta algorithm with a survival random forest model (an example output from the algorithm is provided in the Appendix by Figure B.7.1) where the variables coding for these events will be predictors.
- Boruta algorithm applied at each time point with failure up to current time point as response. A graphical representation of feature importance vs time will be generated similar to the one provided in the Appendix by Figure B.7.2
- Kramer's V evaluated at each time point and represented as a function of time (which will require categorization of continuous variables, to be performed *ad hoc*). A graphical representation of pairwise feature association Kramer's V vs time, similar to the one provided for the Boruta algorithm output represented in he Appendix by Figure B.7.2 will be provided.

Based on the outcome of these exploratory steps, models might be used to investigate further the relationship between these variables and indwell time.

#### 5.2.3.2 Flush pressure profile

Manual flush variability will be evaluated using duration of flush and characteristics of Flush pressure profile obtained on in-line pressure measurements. They will be comprised of:

- Peak pressure
- Flush duration (sec.)

For each of these characteristics, summary statistics by indwell time considered as a discrete variable (0, 6, 24, 30, 48, 54, 72 hours) and longitudinal line and bar plots will be generated on average for continuous and by proportion for categorical responses, respectively.

Lineplots will be similar to the example provided for cfHb in Figure B.3.2 and bar plots will be similar to the example provided for Haemolysis occurrence in Figure B.4.1, both represented in Appendix B.

Relationship between the occurrence of these events will be investigated using the Boruta algorithm with a survival random forest model (an example output from the algorithm is provided in the Appendix by Figure B.7.1) where the variables coding for these events will be predictors.

Based on the outcome of the Boruta algorithm, models might be used to investigate further the relationship between these variables and indwell time.

#### 5.2.4 General Considerations

- For categorical data, count and percentage with 95% confidence interval will be calculated.
- For continuous data, average, standard error, 95% confidence interval, median, inter-quartiles, minimum and maximum will be provided.
- p-values less than 0.05 will be considered statistically significant. Multiple comparisons adjustments (Tukey's or Sydak's) will be made when appropriate
- Importance of factors/variables might be evaluated using machine learning tools such as the Boruta algorithm (random forest all-relevant approach)



- Whenever possible, effects of the following covariates will be investigated: gender, age and BMI
- Initially, all factors/variables will be included into the model as well as any two-way/three-way interactions.
- Variables or interactions which are not significant (p-value < 0.05) will be removed from the final model. Models adjusted with significant effects (and significant interactions if any) will be used for analysis whenever possible.
- Use of models will be preferred to non-parametric tests whenever possible.
- Residual plots for each model will be drawn and reviewed to ensure there are no systematic patterns.
- Transformation of response and/or explanatory variables will be investigated whenever modeling assumptions are not satisfied.

#### 5.2.5 Approaches and Analyses for Missing Data and Other Data Issues

Missing data will not be imputed and will be considered missing for data analysis, resulting in a possible reduced sample size.



## 6 Summary of General Study Data

#### 6.1 Subject Disposition

Participants will be provided the PISCF and once informed, written consent is provided they will be enrolled into the study. Participants will then be screened to ensure they meet the inclusion criteria and do not meet any of the exclusion criteria. Subsequently, participants who are identified as suitable for the study will be provided a unique participant code. The number of participants enrolled and those that failed screening will be recorded. For those that participate in the study, the stage that they reach will also be recorded (e.g., interventional visit 2, as depicted in Figure 6.1.1). For those that participate in the study and drop out, individual responses will be asked to be provided and recorded. Population membership (ITT, PP, etc.) is provided in section 4.1.



Figure 6.1.1: Skeleton flow diagram depicting participant disposition



#### 6.2 Protocol Deviations

Specific protocol deviations are listed below and categorized as either a major deviation (i.e., data to be excluded) or minor (i.e., data to be included).

#### 6.2.1 Major deviations

- Failure to attend: If a participant fails to attend two subsequent visits (e.g. interventional visits 2 & 3), the individual data collected from the participant will be excluded.
- Suspicion of tampering: If it is suspected that the participant has tampered with their PIVCs, as evidenced by breakage of the anti-tampering device, leakage from the extension, perforated dressing the data collected from the participant will be excluded.
- Insertion of alternate gauge PIVCs: Data will be excluded from participants where, in the unanticipated circumstance, a 20G PIVC has been inserted into one arm (e.g., left) of the participant and a 22G PIVC has been inserted into the other arm (e.g., right). Participants will be asked to re-enroll and re-consent after a period of 2 weeks.
- Insertion of identical length PIVCs: Data will be excluded from participants where, in the unanticipated circumstance, two PIVCs of the same length are inserted into the participant regardless of the gauge. Participants will be asked to re-enroll and re-consent after a period of 2 weeks.
- Contraction of a common cold/respiratory infection: If a participant contracts a common cold/respiratory infection during their interventional visit, the individual data collected from that participant will be excluded and they will be removed from the study.

#### 6.2.2 Minor deviations

- Incorrect order for collection of blood: The order in which blood is collected into two alternate size vacutainers (2mL and 6 mL) will be randomized. In the unanticipated circumstance whereby the order of blood collection is incorrect, the data will be included and analyzed "as treated".
- Incorrect order for PIVC insertion: The order in which the PIVCs are inserted into the arm will be randomized. In the unanticipated circumstance whereby the order of PIVC insertion is incorrect, the data will be included and analyzed "as treated".
- Incorrect allocation of PIVC length: The alternate PIVC lengths will be randomized to the participants arms. In the unanticipated circumstance whereby allocation of PIVC length is incorrect (e.g., the 20G 1.0 inch PIVC is inserted into the participant's right arm when it was intended for the participant's left arm), the data will be included and analyzed "as treated".

## 6.3 Demographics and Baseline Variables

Demographic variables will include all medical history questionnaire responses, and each of the following variables at time of intervention:

- Age
- Height
- Weight
- Resting blood pressure
- Gender
- BMI
- Menstrual cycle phase (women only)

Table A.1.1 provides an example of demographic variables summary table, per study group and overall.

Baseline variables will include all sonographic data prior to PIVC insertion and cfHb collected via



venipuncture. Tables A.3.1 and A.3.2 provide examples of baseline variables summary table, per study group and overall, including blood analysis.

#### **6.4** Concurrent Illnesses and Medical Conditions

This study does not aim to recruit individuals with current illnesses. However, in the opinion of the primary investigator and or associated medical opinion, a participant with specific conditions that may not affect blood coagulation and bleeding risk may be considered for inclusion. A list of some illnesses and medical conditions that would result in exclusion and/or may be considered acceptable are indicated below. Please note, specific coding for medical conditions is based upon the International Classification of Diseases (ICD version 11, https://icd.who.int/browse11/l-m/en). Searching the parent classification will provide examples of specific conditions. For brevity, we have provided only codes and descriptions for ICD-11\_03 (Disease of the blood or blood-forming organs).

Table 6.4.1: List of medical conditions that will exclude participants from participating in this trial

| Parent Classification | Code/s | Description |
|---|---|---|
| ICD-11_01 | | Any and all infections will exclude volunteers from participating |
| ICD-11_02 | _ | Any and all neoplasms will exclude volunteers from participating |
| ICD-11_03 | 3B10 | Hereditary factor VIII deficiency |
| Disease of the blood or | 3B11 | Hereditary factor IX deficiency |
| blood-forming organs | 3B12 | Von Willebrand disease |
| | 3B13 | Haemophilia C |
| | 3B14 | Other inherited coagulation factor deficiency with bleeding tendency |
| | 3B15 | Inherited coagulation factor deficiency without bleeding tendency |
| | 3B20 | Disseminated intravascular coagulation |
| | 3B21 | Haemorrhagic disorder due to circulating anticoagulants and coagulation factors |
| | 3B22 | Acquired haemophilia |
| | 3B50 | Inherited fibrinolytic defects |
| | 3B51 | Acquired fibrinolytic defects |
| | 3B60 | Non-thrombocytopenic purpura |
| | 3B61 | Thrombophilia |
| | 3B62 | Qualitative platelet defects |
| | 3B63 | Thrombocytosis |
| | 3B64 | Thrombocytopenia |
| | 3B65 | Thrombotic microangiopathy, not elsewhere classified |
| | 3B80 | Congenital disorders of spleen |
| | 3B81 | Acquired disorders of spleen |
| ICD-11_04 | _ | Any and all diseases of the immune system will exclude volunteers from participating |
| ICD-11_05 | _ | Any and all endocrine, nutritional or metabolic diseases will exclude volunteers from partic- |
| | | ipating |
| ICD-11_06 | _ | Specifically, the following codes will be excluded: 6A20-6A25, 6A40, 6A40, 6A60-6A62, 6A71- |
| | | 6A73, 6B01-6B03, 6B06, 6B23, 6B25, 6B40-6B43, 6B61-6B66, 6B80-6B85, 6C00, 6C01, 6C20, 6C01, 6C01, 6C02, 6C01, 6C |
| | | 6C21, 6C40-6C4H, 6C50, 6C51, 6C70-6C73, 6C90, 6C91, 6D30-6D36, 6D50, 6D51, 6D70- |
| | | 6D72, 6D80-6D86, 6E40, 6E60-6E-69. The inclusion of participants with mental, behavioural |
| | | or neurodevelopmental disorders not specifically listed here (including sub-classifications) will |
| | | be decided by the PI on a 'case-by-case' basis. |
| ICD-11_07 | _ | Any and all sleep-wake disorders will exclude volunteers from participating |
| ICD-11_08 | | Specifically, the following codes will be excluded: 8A00-8A07, 8A20-8A23, 8A40-8A46, 8A60- |
| | | 8A68, 8B00-8B03, 8B10, 8B11, 8B20-8B26, 8B40-8B44, 8B60-8B62, 8B85, 8B86, 8B88, 8B90- |
| | | 8B94, 8C00-8C03, 8C10-8C12, 8C20, 8C21, 8C60-8C62, 8C70-8C78, 8C80-8C84, 8D20-8D23, |
| | | 8D40-8D44, 8D60-8D68, 8D80-8D8C, 8E00-8E03, 8E20-8E22, 8E40-8E4A, 8E60-8E66. The |
| | | inclusion of participants with diseases of the nervous system not specifically listed here (in- |
| | | cluding sub-classifications) will be decided by the PI on a 'case-by-case' basis. |
| ICD-11_09 | _ | Specifically, the following codes will be excluded: 9A01, 9A02, 9A10, 9A11, 9A21-9A23, |
| | | 9A60, 9A61, 9A71, 9A73, 9A76, 9A80-9A83, 9A91, 9A96, 9B50, 9B51, 9B63, 9B65, 9B66, |
| | | 9B71-9B78, 9B82, 9B83, 9C20-9C22, 9C60, 9C61, 9D20-9D25. The inclusion of participants |
| | | with diseases of the visual system not specifically listed here (including sub-classifications) |
| | | will be decided by the PI on a 'case-by-case' basis. |
| ICD-11_10 | | Specifically, the following codes will be excluded: AA00-AA04, AA90, AA91, AB00, AB01, |
| | | AB10-AB1B, AB30-AB36, AB53, AB70, AB71, AB90-AB93. The inclusion of partici- |
| | | pants with diseases of the ear or mastoid process not specifically listed here (including sub- |
| | | classifications) will be decided by the PI on a 'case-by-case' basis. |
| | | , |



| ICD-11_11 | _ | Any and all diseases of the circulatory system will exclude volunteers from participating |
|---|---|---|
| ICD-11_12 | _ | Any and all diseases of the respiratory system will exclude volunteers from participating |
| ICD-11_13 | _ | Any and all diseases of the digestive system will exclude volunteers from participating |
| ICD-11_14 | _ | Specifically, the following codes will be excluded: EA00, EA10-EA12, EA20, EA50, EA51, EA60, EA89, EB00, EB04, EB05, EB10-EB31, EB40-EB44, EB50, EB51, EB61, EB90, EC20, EC30-EC33, EC40, EC90-EC92, ED00-ED02, ED30, ED50-ED56, ED60, ED62, EE00, EE02, EE20, EE21, EE40, EE41, EE50, EE70, EE80, EE81, EE90, EE91, EF20, EF30, EF31, EF40, EF50, EF60, EG00-EG02, EH77, EH90-EH93, EJ10, EJ30, EJ70, EJ71, EK00-EK02, EK10-EK12, EK70, EL10, EL50-EL54, EL60-EL62, EL70-EL73, EL80. The inclusion of participants with diseases of the skin not specifically listed here (including sub-classifications) will be decided by the PI on a 'case-by-case' basis. |
| ICD-11_15 | _ | Specifically, the following codes will be excluded: FA10-FA13, FA-FA27, FA36, FA70-FA72, FA80-FA85, FA90-FA92, FB00, FB10, FB30-FB33, FB40-FB43, FB50-FB56, FB80-FB86, FC01. The inclusion of participants with diseases of the musculoskeletal system or connective tissue not specifically listed here (including sub-classifications) will be decided by the PI on a 'case-by-case' basis. |
| ICD-11_16 | | Specifically, the following codes will be excluded: GA00-GA07, GA20-GA23, GA30, GA91, GB07, GB08, GB21, GB23, GB40-GB42, GB50-GB59, GB60, GB61, GB70, GB71, GB80-GB83, GB90, GC00-GC08. The inclusion of participants with diseases of the genitourinary system—not specifically listed here (including sub-classifications) will be decided by the PI on a 'case-by-case' basis. |
| ICD-11_17 | _ | None to consider |
| ICD-11_18 | _ | Any and all conditions associated with pregnancy, childbirth or puerpium will exclude vol-<br>unteers from participating |
| ICD-11_19 | _ | Not applicable |
| ICD-11_20 | | Specifically, the following codes will be excluded: LA00-LA07, LA70-LA77, LA80-LA8G, LA90, LB00, LB20-LB22, LB30, LB31, LB72-LB74, LB90-LB92, LB96, LB96, LB99, LC00-LC02, LC20, LC50-LC52, LC60, LC80, LD20, LD23, LD24, LD26-LD29, LD2C-LD2H, LD40-LD47, LD90. The inclusion of participants with developmental anomalies not specifically listed here (including sub-classifications) will be decided by the PI on a 'case-by-case' basis. |
| ICD-11_21 | | Any and all symptoms, signs, or clinical findings not elsewhere classified will exclude volunteers from participating |
| ICD-11_22 | _ | Any injury, poisoning or certain other consequences of external causes except for NC50 and ND10, will exclude volunteers from participating |
| ICD-11_23 | | Not applicable |

## 6.5 Prior and Concurrent Medications

This study does not aim to recruit individuals who are regularly taking medications. However, in the opinion of the primary investigator and or associated medical opinion, a participant taking medications that may not affect blood coagulation and bleeding risk may be considered for inclusion. A list of some drug classes and example drugs that would result in exclusion and/or may be considered acceptable are indicated below.

Please note, specific coding for drugs, based upon the ATC/DDD Index 2020 (https://www.whocc.no/atc\_ddd\_index/) are listed to provide some specific examples. Searching the drug classes can provide specific examples. Specific examples of drugs within the B01A Antithrombotic Agents class are given for example.

Table 6.5.1: List of current drug use resulting in exclusion (1/2)

| D 01 | | | |
|---|---|---|---|
| Drug Class | Drug Class Description | $\operatorname{Drug}$ | Description |
| B01AA | Vitamin K Antagonists | B01AA03 | Warfarin |
| B01AB | Heparin Group | B01AB01 | Heparin |
| B01AC | Platelet Aggregation Inhibitors | B01AC04 | Clopidogrel |
| | Excl. Heparin | | |
| | | B01AC06 | Acetylsalicylic Acid |
| | | B01AC16 | Eptifibatide |
| | | B01AC24 | Ticagrelor |
| B01AD | Enzymes | B01AD01 | Streptokinase |
| | B01AA<br>B01AB<br>B01AC | B01AA Vitamin K Antagonists B01AB Heparin Group B01AC Platelet Aggregation Inhibitors Excl. Heparin | B01AA |



| | | B01AD04 | Urokinase |
|-------|-----------------------------|---------|--------------|
| | | B01AD11 | Tenecteplase |
| B01AE | Direct Thrombin Inhibitors | B01AE06 | Bivalirudin |
| B01AF | Direct Factor Xa Inhibitors | B01AF01 | Rivaroxaban |
| B01AX | Other Antithrombotic Agents | B01AX01 | Defibrotide |



Table 6.5.2: List of current drug use resulting in exclusion (2/2)

| Class | Parent Classification | Drug Class | Drug Class Description |
|---|---|---|---|
| J01 | J01A | - Ling Class | Drug Class Description |
| Antibacterials for Systemic<br>Use | Tetracyclines | _ | |
| Ose | J01B | _ | |
| | Amphenicols | | |
| | J01C | _ | |
| | Beta-lactam Antibacterials, Penicillins | | |
| | J01D | _ | |
| | Other Beta-lactam Antibacterials | | |
| | m J01E | - | |
| | Sulphonamides and Trimethoprim | | |
| | J01F | _ | |
| | Macrolides, Lincosamides and Streptogramins J01G | _ | |
| | Aminoglycoside Antibacterials | | |
| | J01M | _ | |
| | Quinoline Antibacterials | | |
| | J01R | _ | |
| | Combinations of Antibacterials | | |
| | J01X | - | |
| | Other Antibacterials | | |
| J02 | J02A | J02AA | Antibiotics |
| Antimycotics for systemic<br>Use | Antimycotics for Systemic Use | J02AB | Imidazole Derivatives |
| OSC | | m J02AC $ m J02AX$ | Triazole Derivatives Other Antimycotics for Systemic Use |
| J04 | m J04A | 302AA | Other Antimycotics for Systemic Ose |
| Antimycobacterials | Drugs for Treatment of Tuberculosis | | |
| | J04B | _ | |
| | Drugs for Treatment of Lepra | | |
| J05 | J05A | - | |
| Antivirals for Systemic Use | Direct Acting Antivirals | | |
| J06 | J06A | - | |
| Immune Sera and Immunoglobulins | Immune Sera | | |
| | J06B | _ | |
| | Immunoglobulins | | |
| J07 | J07A | _ | |
| Vaccines | Bacterial Vaccines | | |
| | J07B | - | |
| | Viral Vaccines | | |
| | J07C | - | |
| | Plant Alkaloids | | |
| | J07X | - | |
| | Other Vaccines | | |
| L01 | L01A | - | |
| Antineoplastic and Immunomodulating Agents | Alkylating Agents | | |
| | L01B | - | |
| | Antimetabolites | | |
| | L01C | - | |
| | Plant Alkaloids and Other Natural Products | | |
| | L01D | - | |
| | Cytotoxic Antibiotics and Related Substances<br>L01X | | |
| | Other Antineoplastic Agents | - | |
| L04 | L04A | L04AA | Selective Immunosupressants |
| Immunosupressants | Immunosupressants | L04AX | Other Immunosupressants |
| | | | 5 IIIIII alloo aprobballoo |

An example of other drug classes which may not result in exclusion, but will trigger deeper investigation



for their effect on platelet function/thrombosis is provided in Table 6.5.3.

Table 6.5.3: List of current drug use trigerring deeper investigation for their effect on platelet function/thrombosis

| Class | Parent Classification | Drug Class | Drug Class Description |
|---|---|---|---|
| G03 | G03A | G03AA | Progestogens and Estrogens, |
| | | | fixed combinations |
| Sex Hormones and Modulators | Hormonal Contraceptives for | | |
| of the Genital System | Systemic Use | | |
| | | G03AB | Progestogens and Estrogens, |
| | | | sequential preparations |
| | | G03AC | Progestogens |
| N02 | N02A | N02AA | Natural Opium Alkaloids |
| Analgesics | Opioids | N02AB | Phenylpiperidine Derivatives |
| | | N02AC | Diphenylpropylamine Derivatives |
| | | N02AD | Benzomorphan Derivatives |
| | | N02AE | Oripavine Derivatives |
| | | N02AF | Morphinan Derivatives |
| | | N02AG | Opioids in Combination with |
| | | | Antispasmodics |
| | | N02AJ | Opioids in Combination with |
| | | | Non-opioid Analgesics |
| | | N02AX | Other Opioids |
| | N02B | N02BA | Salicylic Acid and Derivatives |
| | Other Analgesics and Antipyretics | N02BB | Pyrazolones |
| | | N02BE | Anilides |
| | N02C | N02CA | Ergot Alkaloids |
| | Antimigraine Preparations | N02CB | Corticosteroid Derivatives |
| | | N02CC | Selective Serotonin (5HT1) |
| | | | Agonists |
| | | N02CD | Calcitonin Gene-related Pep- |
| | | | tide (CGRP) Antagonists |
| | | N02CX | Other Antimigraine Prepara- |
| | | | tions |

## 6.6 Device Failure, Malfunctions and Defects

PIVC failure in the current study is defined as:

- 1. An inability to flush or collect blood through the PIVC
- 2. The removal of the PIVC based on medical doctor's assessment of an AE

A device rescue decision tree (see Appendix 16.5 of the study protocol) will be utilized to identify if the PIVC has failed.

## 7 Safety Analysis

Sufficient detail on summarizing safety data, e.g., information on severity, expectedness, and causality; details of how adverse events are coded or categorized; how adverse event data will be analyzed is provided in a separate document (i.e., a safety management plan).

## 8 Interim Analysis Plan

No interim analysis has been planned.



## 9 References

- [1] R Core Team. R: A Language and Environment for Statistical Computing. R Foundation for Statistical Computing, Vienna, Austria, 2016. URL https://www.R-project.org/.
- [2] Miron B. Kursa and Witold R. Rudnicki. Feature selection with the Boruta package. *Journal of Statistical Software*, 36(11):1–13, 2010. URL http://www.jstatsoft.org/v36/i11/.



## 10 SAP Revision History

| Version Number | Rationale for Change | Section or Page Affected | Description of Change |
|---|---|---|---|
| 1.0 | Original SAP | | |



## 11 Appendix

## A Tables

## A.1 Demographics

Table A.1.1: Numerical Summary of Subjects Demographics, per Group (i.e. Gauge) and Overall

| Characteristic | 20G | 22G | Overall |
|--------------------------|----------------|----------------|----------------|
| Age (years) | | | |
| Mean | 42.35 | 39.87 | 41.11 |
| 95% Mean CI | 37.42, 47.07 | 34.77, 44.98 | 37.51, 44.70 |
| Median | 45.15 | 39.45 | 42.15 |
| $\operatorname{SD}$ | 11.22 | 12.14 | 11.61 |
| Min, Max | 24.2, 56.3 | 23.9, 57.4 | 23.9, 57.4 |
| Total Count | 20 | 20 | 40 |
| Gender | | | |
| F | 11 (55.0%) | 9 (45.0%) | 20 (50.0%) |
| M | 9 (45.0%) | 11(55.0%) | 20 (50.0%) |
| Total | 20 | 20 | 40 |
| Ethnicity | | | |
| Non Hispanic / Latino | 18 (90.0%) | 19 (95.0%) | 37 (92.5%) |
| Hispanic / Latino | 2 (10.0%) | 1 (5.0%) | 3 (7.5%) |
| Total | 20 | 20 | 40 |
| Race | | | |
| Asian | 6 (30.0%) | 8 (40.0%) | 14 (35.0%) |
| Other | 7 (35.0%) | 6 (30.0%) | 13 (32.5%) |
| White / Caucasian | 7 (35.0%) | 6 (30.0%) | 13 (32.5%) |
| Total | 20 | 20 | 40 |
| Height (cm) | | | |
| Mean | 166.06 | 168.64 | 167.35 |
| 95% Mean CI | 161.10, 171.26 | 163.55, 173.65 | 163.63, 171.10 |
| Median | 161.05 | 168.20 | 166.65 |
| $\operatorname{SD}$ | 12.09 | 11.78 | 11.85 |
| Min, Max | 151.2, 185.6 | 150.4, 188.6 | 150.4, 188.6 |
| Total Count | 20 | 20 | 40 |
| Weight (kg) | | | |
| Mean | 67.92 | 76.78 | 72.34 |
| 95% Mean CI | 63.44, 72.27 | 73.23, 80.32 | 69.18, 75.43 |
| Median | 72.50 | 76.10 | 74.75 |
| $\operatorname{SD}$ | 10.41 | 8.34 | 10.34 |
| Min, Max | 52.8, 81.6 | 63.5, 88.7 | 52.8, 88.7 |
| Total Count | 20 | 20 | 40 |
| BMI (kg/m <sup>2</sup> ) | | | |
| Mean | 22.40 | 22.90 | 22.65 |
| 95% Mean CI | 21.25, 23.55 | 21.85, 24.00 | 21.88, 23.45 |
| Median | 23.00 | 23.50 | 23.00 |
| $\operatorname{SD}$ | 2.68 | 2.55 | 2.60 |
| Min, Max | 18, 27 | 19, 27 | 18, 27 |
| Total Count | 20 | 20 | 40 |

## A.2 Family Medical History

Table A.2.1: Numerical Summary of Familiy Medical History, per Group (i.e. Gauge) and Overall

| v v | 0 / L | • ( | 0 / |
|---|---|---|---|
| Characteristic | 20G | 22G | Overall |
| Blood Disorder or Bleeding or Clotting Problem | | | |
| No | $20 \ (100.0\%)$ | 18 (90.0%) | 38 (95.0%) |
| Yes | 0 ( 0.0%) | 2(10.0%) | 2 ( 5.0%) |
| Total | 20 | 20 | 40 |



 $\hbox{ Table A.2.1: Numerical Summary of Familiy Medical History, per Group (i.e. \ Gauge) and \ Overall \ continued$ 

| Characteristic | 20G | 22G | Overall |
|---|---|---|---|
| Cancer | | | |
| No | 19 (95.0%) | 19 (95.0%) | 38 (95.0%) |
| Yes | 1 (5.0%) | 1 (5.0%) | 2(5.0%) |
| Total | 20 | 20 | 40 |
| Heart Disease | | | |
| No | $20 \ (100.0\%)$ | $20 \ (100.0\%)$ | 40 (100.0%) |
| Yes | 0 ( 0.0%) | 0 ( 0.0%) | 0 ( 0.0%) |
| Total | 20 | 20 | 40 |
| High Blood Pressure (Hypertension) | | | |
| No | 13~(65.0%) | 19 (95.0%) | 32 (80.0%) |
| Yes | 7 (35.0%) | 1 (5.0%) | 8 (20.0%) |
| Total | 20 | 20 | 40 |
| Diabetes Type 2 | | | |
| No | 19 (95.0%) | 14 (70.0%) | 33 (82.5%) |
| Yes | 1 (5.0%) | 6 (30.0%) | 7 (17.5%) |
| Total | 20 | 20 | 40 |

## A.3 Baseline Characteristics

Table A.3.1: Numerical Summary of Baseline PIVC Characteristics, per Group (i.e. Gauge) and Overall

| Characteristic | 20G | 22G | Overall |
|---|---|---|---|
| Tip Position Mid-Stream | | | |
| Yes | 16 (80.0%) | 15~(75.0%) | $31\ (77.5\%)$ |
| No | 4(20.0%) | 5(25.0%) | 9(22.5%) |
| Total | 20 | 20 | 40 |
| Tip Position Well Contact | | | |
| No | 16 (80.0%) | 17 (85.0%) | 33~(82.5%) |
| Yes | 4(20.0%) | 3(15.0%) | 7 (17.5%) |
| Total | 20 | 20 | 40 |
| Blood Flow Velocity (cm/sec) | | | |
| Mean | 161.94 | 161.86 | 161.90 |
| 95% Mean CI | 159.06, 164.96 | 159.05, 164.73 | 159.86, 163.97 |
| Median | 160.97 | 162.27 | 161.69 |
| SD | 6.90 | 6.61 | 6.67 |
| Min, Max | 150.46, 173.71 | 150.97, 173.28 | 150.46, 173.71 |
| Total Count | 20 | 20 | 40 |
| Catheter-to-Vein ratio | | | |
| Mean | 38.70 | 35.92 | 37.31 |
| 95% Mean CI | 36.95, 40.42 | 34.27, 37.56 | 36.02, 38.61 |
| Median | 38.88 | 35.06 | 36.93 |
| SD | 4.13 | 3.91 | 4.21 |
| Min, Max | 32.11, 44.91 | 30.23, 42.67 | 30.23, 44.91 |
| Total Count | 20 | 20 | 40 |

 $\begin{tabular}{ll} Table A.3.2: Numerical Summary of Baseline Venipuncture Blood Analysis, per Group (i.e. Gauge) and Overall \\ \end{tabular}$ 

| Tube Volume | Characteristic | 20G | 22G | Overall |
|---|---|---|---|---|
| 2mL | cfHb (mg/dL) | | | |
| | Mean | 199.31 | 200.93 | 200.12 |
| | 95% Mean CI | 175.48, 222.22 | 174.31, 228.18 | 182.19, 218.30 |
| | Median | 201.03 | 199.82 | 199.82 |
| | $\operatorname{SD}$ | 53.78 | 64.40 | 58.57 |
| | Min, Max | 56.99, 324.24 | 111.27, 317.8 | 56.99, 324.24 |
| | Total Count | 20 | 20 | 40 |



 $\begin{tabular}{ll} Table A. 3.2: Numerical Summary of Baseline Venipuncture Blood Analysis, per Group (i.e. Gauge) and Overall continued \\ \end{tabular}$ 

| Tube Volume | Characteristic | 20G | 22G | Overall |
|---|---|---|---|---|
| | Haemolysis - AU480 (Yes/No) | | | |
| | No | 10 (50.0%) | 10 (50.0%) | 20 (50.0%) |
| | Yes | 10 (50.0%) | 10 (50.0%) | 20 (50.0%) |
| | Total | 20 | 20 | 40 |
| | Haemolysis - Visual (Yes/No) | | | |
| | Yes | 14 (70.0%) | 12 (60.0%) | 26 (65.0%) |
| | No | 6 (30.0%) | 8 (40.0%) | 14 (35.0%) |
| | Total | 20 | 20 | 40 |
| | Blood Draw Fill Time (sec) | | | |
| | Mean | 39.48 | 39.15 | 39.31 |
| | 95% Mean CI | 37.86, 41.08 | 37.41, 40.86 | 38.10, 40.51 |
| | Median | 39.40 | 39.92 | 39.74 |
| | $\operatorname{SD}$ | 3.83 | 4.06 | 3.90 |
| | Min, Max | 32.77, 46.32 | 32.06, 46.4 | 32.06, 46.4 |
| | Total Count | 20 | 20 | 40 |
| 6mL | cfHb (mg/dL) | | | |
| | Mean | 194.94 | 200.96 | 197.95 |
| | 95% Mean CI | 174.19, 215.28 | 178.16, 223.07 | 182.86, 213.25 |
| | Median | 212.88 | 193.48 | 207.24 |
| | $\operatorname{SD}$ | 47.91 | 52.64 | 49.77 |
| | Min, Max | 86.01, 275.98 | 103.33, 311.35 | 86.01, 311.35 |
| | Total Count | 20 | 20 | 40 |
| | Haemolysis - AU480 (Yes/No) | | | |
| | Yes | 12 (60.0%) | 9 (45.0%) | 21 (52.5%) |
| | No | 8 (40.0%) | 11(55.0%) | 19 (47.5%) |
| | Total | 20 | 20 | 40 |
| | Haemolysis - Visual (Yes/No) | | | |
| | Yes | 13 (65.0%) | 13 (65.0%) | 26 (65.0%) |
| | No | 7 (35.0%) | 7 (35.0%) | 14 (35.0%) |
| | Total | 20 | 20 | 40 |
| | Blood Draw Fill Time (sec) | | | |
| | Mean | 99.94 | 101.73 | 100.83 |
| | 95% Mean CI | 97.33, 102.41 | 98.61, 105.01 | 98.85, 102.95 |
| | Median | 101.04 | 100.15 | 100.15 |
| | $\operatorname{SD}$ | 5.98 | 7.49 | 6.75 |
| | Min, Max | 86.61, 108.96 | 91.1, 116.4 | 86.61, 116.4 |
| | Total Count | 20 | 20 | 40 |


#### A.4 Indwell Time

Table A.4.1: Numerical Summary of Subjects Indwell Time in hours, per Device Configuration (Gauge and Length) and Overall

| | <del>-</del> | | | | |
|---|---|---|---|---|---|
| Characteristic | BD Nexiva (22G | BD Nexiva (22G | BD Nexiva (20G | BD Nexiva (20G | Overall |
| | x 1 inch) | x 1.75 inch) | x 1 inch) | x 1.75 inch) | |
| Indwell Time (Hours) | | | | | |
| Mean | 44.76 | 55.84 | 59.72 | 69.82 | 57.54 |
| 95% Mean CI | 36.08, 53.42 | 45.68, 64.78 | 52.74, 65.55 | 68.08, 71.24 | 53.19, 61.60 |
| Median | 42.84 | 66.22 | 64.09 | 72.00 | 66.97 |
| $\operatorname{SD}$ | 20.38 | 22.59 | 14.76 | 3.83 | 18.97 |
| Min, Max | 9.4, 72 | 0.07, 72 | 15.76, 72 | 58.6, 72 | 0.07, 72 |
| Total Count | 20 | 20 | 20 | 20 | 80 |

Table A.4.2: Proportional Hazard Ratios computed from Cox Proportional Hazards model for Indwell time

| | HR(95%CI) | P(Wald's test) | P(LR-test) |
|---|---|---|---|
| device: ref.=BD Nexiva (22G x 1 inch) | | | 0.002 |
| BD Nexiva (22G x 1.75 inch) | $0.6 \ (0.28, 1.26)$ | 0.175 | |
| BD Nexiva (20G x 1 inch) | 0.57(0.27,1.2) | 0.141 | |
| BD Nexiva (20G x 1.75 inch) | $0.2\ (0.08, 0.49)$ | < 0.001 | |



#### A.5 Indwell Failure Mode

Table A.5.1: Failure Modes Count Overall

| Failure Mode | Flush | Draw (2mL) | Draw (6mL) |
|--------------------------|-------|------------|------------|
| Unsecure Luer Connection | 2 | 0 | 1 |
| Locked Clamps | 2 | 0 | 0 |
| Catheter Dislodgement | 5 | 0 | 0 |
| Catheter Kinking | 2 | 2 | 0 |
| Vasospasm | 0 | 0 | 0 |
| Thrombus | 24 | 10 | 7 |
| Infiltration | 2 | 0 | 0 |
| Other | 9 | 0 | 1 |

A list of the failure modes available in the free form text field describing the "Other" category will be provided.

Table A.5.2: Failure Modes Count Per Device Configuration

| Device | Failure Mode | Flush | Draw (2mL) | Draw (6mL) |
|---|---|---|---|---|
| BD Nexiva (22G x 1 inch) | Luer Connection | 0 | 0 | 0 |
| | Clamp | 1 | 0 | 0 |
| | Tube Kinking | 0 | 0 | 0 |
| | Dislodgement | 0 | 0 | 0 |
| | Catheter Kinking | 1 | 0 | 0 |
| | Vasospasm | 0 | 0 | 0 |
| | Thrombus | 9 | 2 | 2 |
| | Infiltration | 0 | 0 | 0 |
| | Other | 5 | 0 | 0 |
| BD Nexiva (22G x 1.75 inch) | Luer Connection | 0 | 0 | 1 |
| | Clamp | 0 | 0 | 0 |
| | Tube Kinking | 0 | 0 | 0 |
| | Dislodgement | 2 | 0 | 0 |
| | Catheter Kinking | 0 | 0 | 0 |
| | Vasospasm | 0 | 0 | 0 |
| | Thrombus | 6 | 1 | 2 |
| | Infiltration | 1 | 0 | 0 |
| | Other | 2 | 0 | 0 |
| BD Nexiva (20G x 1 inch) | Luer Connection | 1 | 0 | 0 |
| | Clamp | 1 | 0 | 0 |
| | Tube Kinking | 0 | 0 | 0 |
| | Dislodgement | 2 | 0 | 0 |
| | Catheter Kinking | 1 | 1 | 0 |
| | Vasospasm | 0 | 0 | 0 |
| | Thrombus | 7 | 3 | 3 |
| | Infiltration | 1 | 0 | 0 |
| | Other | 1 | 0 | 1 |
| BD Nexiva (20G x 1.75 inch) | Luer Connection | 1 | 0 | 0 |
| | Clamp | 0 | 0 | 0 |
| | Tube Kinking | 0 | 0 | 0 |
| | Dislodgement | 1 | 0 | 0 |
| | Catheter Kinking | 0 | 1 | 0 |
| | Vasospasm | 0 | 0 | 0 |
| | Thrombus | 2 | 4 | 0 |
| | Infiltration | 0 | 0 | 0 |
| | Other | 1 | 0 | 0 |

### A.6 Indwell Failure Mode Per Day

Table A.6.1: Failure Modes Count Overall Per Day

| | | | | | | | | · | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Failure Mode | Day 1: | Day 1: | Day 1: | Day 2: | Day 2: | Day 2: | Day 3: | Day 3: | Day 3: | Day 4: | Day 4: | Day 4: |
| | Flush | Blood | Blood | Flush | Blood | Blood | Flush | Blood | Blood | Flush | Blood | Blood |
| | | Draw | Draw | | Draw | Draw | | Draw | Draw | | Draw | Draw |
| | | (2mL) | (6mL) | | (2mL) | (6mL) | | (2mL) | (6mL) | | (2mL) | (6mL) |
| Luer Connection | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 |
| Clamp | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 |
| Tube Kinking | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Dislodgement | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 |
| Catheter Kinking | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 |
| Vasospasm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Thrombus | 2 | 1 | 1 | 6 | 2 | 0 | 9 | 2 | 2 | 7 | 5 | 4 |
| Infiltration | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 |
| Other | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 1 |



Table A.6.2: Failure Modes Count Per Device Configuration

| Device | Failure Mode | Day 1:<br>Flush | Day 1:<br>Blood | Day 1:<br>Blood | Day 2:<br>Flush | Day 2:<br>Blood | Day 2:<br>Blood | Day 3:<br>Flush | Day 3:<br>Blood | Day 3:<br>Blood | Day 4:<br>Flush | Day 4:<br>Blood | Day 4:<br>Blood |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Flush | Blood<br>Draw | Blood<br>Draw | Flush | Blood<br>Draw | | Flush | | Blood<br>Draw | Flush | | Blood<br>Draw |
| | | | (2mL) | (6mL) | | (2mL) | Draw<br>(6mL) | | $\frac{\text{Draw}}{(2\text{mL})}$ | (6mL) | | $\frac{\text{Draw}}{(2\text{mL})}$ | (6mL) |
| DD Nasier (22C 1 in dr) | Catheter Kinking | 4 | 0 | , | 0 | , , | 0 | 0 | | 0 | 0 | , , | (OIIIL) |
| BD Nexiva (22G x 1 inch) | | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | - | 0 | 0 | 0 |
| | Clamp | 0 | o . | | 0 | 0 | - | 1 | 0 | 0 | 0 | 0 | 0 |
| | Dislodgement | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | Infiltration | 0 | 0 | 0 | 0 | 0 | 0 | U | 0 | 0 | 0 | 0 | 0 |
| | Luer Connection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | Other | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |
| | Thrombus | 2 | 0 | 0 | 5 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 1 |
| | Tube Kinking | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | Vasospasm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| BD Nexiva (22G x 1.75 inch) | Catheter Kinking | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | Clamp | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | Dislodgement | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 |
| | Infiltration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |
| | Luer Connection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
| | Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 |
| | Thrombus | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 1 |
| | Tube Kinking | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | Vasospasm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| BD Nexiva (20G x 1 inch) | Catheter Kinking | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 |
| , | Clamp | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |
| | Dislodgement | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 |
| | Infiltration | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |
| | Luer Connection | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |
| | Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 |
| | Thrombus | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 1 | 1 | 2 | 1 | 2 |
| | Tube Kinking | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | Vasospasm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| BD Nexiva (20G x 1.75 inch) | Catheter Kinking | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 |
| 22 Tem (200 H 11/0 men) | Clamp | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | Ô |
| | Dislodgement | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |
| | Infiltration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | Luer Connection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |
| | Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |
| | Thrombus | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 |
| | Tube Kinking | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 - |
| | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | Vasospasm | U | U | U | U | U | U | U | U | U | U | U | U C |



#### A.7 Failure Remediation

Table A.7.1: Remediation Steps Count Overall

| Step | Flush | Draw (2mL) | Draw (6mL) |
|-------------------------------|-------|------------|------------|
| No remediation | 0 | 0 | 0 |
| Secure Luer | 0 | 0 | 0 |
| Clamp Release | 0 | 0 | 0 |
| Tube Unkink | 0 | 0 | 0 |
| Digital Pressure | 0 | 0 | 0 |
| Dressing Replacement | 0 | 0 | 0 |
| Dressing w/Digital Pressure | 0 | 0 | 0 |
| First tourniquet | 0 | 0 | 0 |
| Tourniquet w/Digital Pressure | 0 | 0 | 0 |
| Heat Pack | 0 | 0 | 0 |
| Heat Pack w/Digital Pressure | 0 | 0 | 0 |
| Second tourniquet | 0 | 0 | 0 |
| Tourniquet w/Digital Pressure | 0 | 0 | 0 |
| Unable to Rescue | 0 | 0 | 0 |

A similar table will be provided detailing counts per Device Configuration.

Table A.7.2: Remediation Characteristics Count per Device Configuration per Day

| Device | Characteristic | Day 1 | Day 2 | Day 3 | Day 4 |
|---|---|---|---|---|---|
| BD Nexiva (22G x 1 inch) | Total Number of Attempts | 0 | 0 | 0 | 0 |
| | No Remediation | 0 | 0 | 0 | 0 |
| | Success with Remediation | 0 | 0 | 0 | 0 |
| | Unsuccessful with Remediation | 0 | 0 | 0 | 0 |
| BD Nexiva (22G x 1.75 inch) | Total Number of Attempts | 0 | 0 | 0 | 0 |
| | No Remediation | 0 | 0 | 0 | 0 |
| | Success with Remediation | 0 | 0 | 0 | 0 |
| | Unsuccessful with Remediation | 0 | 0 | 0 | 0 |
| BD Nexiva (20G x 1 inch) | Total Number of Attempts | 0 | 0 | 0 | 0 |
| | No Remediation | 0 | 0 | 0 | 0 |
| | Success with Remediation | 0 | 0 | 0 | 0 |
| | Unsuccessful with Remediation | 0 | 0 | 0 | 0 |
| BD Nexiva (20G x 1.75 inch) | Total Number of Attempts | 0 | 0 | 0 | 0 |
| | No Remediation | 0 | 0 | 0 | 0 |
| | Success with Remediation | 0 | 0 | 0 | 0 |
| | Unsuccessful with Remediation | 0 | 0 | 0 | 0 |

# A.8 Blood Analysis

Table A.8.1: Numerical Summary of Subjects Blood Analysis, for each time point, per Device Configuration (Gauge and Length) and Vacutainer tube and Overall

| Time<br>Point<br>(hours) | Characteristic | BD Nexiva (22G<br>x 1 inch) - 2mL | BD Nexiva (22G<br>x 1 inch) - 6mL | BD Nexiva (22G<br>x 1.75 inch) -<br>2mL | BD Nexiva (22G<br>x 1.75 inch) -<br>6mL | BD Nexiva (20G<br>x 1 inch) - 2mL | BD Nexiva (20G<br>x 1 inch) - 6mL | BD Nexiva (20G<br>x 1.75 inch) -<br>2mL | BD Nexiva (20G<br>x 1.75 inch) -<br>6mL | Overall |
|---|---|---|---|---|---|---|---|---|---|---|
| 0 | cfHb (mg/dL) | 100.10 | .=0.11 | 101.10 | 1=0.00 | 450.00 | | 110.00 | | |
| | Mean<br>95% Mean<br>CI | $196.10 \\ 171.35, 219.19$ | 178.14<br>158.51, 197.03 | $164.49 \\ 150.93, 178.84$ | 172.33<br>160.06, 184.58 | 172.62 $159.35, 186.12$ | | $149.22 \\ 139.16, 160.00$ | $147.86 \\ 139.67, 155.47$ | 167.59<br>161.88, 173.62 |
| | Median<br>SD | 195.08<br>55.75 | 180.15 $45.54$ | 155.63 $32.54$ | 167.18<br>28.87 | $162.05 \\ 31.76$ | 157.74 $39.52$ | $152.27 \\ 24.26$ | 151.02<br>18.39 | 160.67 $38.54$ |
| | Min, Max | 76.06, 303.33 | 97.93, 260.95 | 108.78, 234.07 | 128.96, 230.49 | 128.66, 228.95 | 103.03, 242.28 | 100.59, 215.9 | 98.15, 179.49 | 76.06, 303.33 |
| | Total<br>Count<br>Haemolysis | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 160 |
| | - AU480<br>(Yes/No) | | | | | | | | | |
| | No | 12 (60.0%) | 14 (70.0%) | 16 (80.0%) | 16 (80.0%) | 14 (70.0%) | 17 (85.0%) | 19 (95.0%) | 20 (100.0%) | 128 (80.0%) |
| | $_{ m Yes}$ $_{ m Total}$ | 8 (40.0%)<br>20 | 6 (30.0%)<br>20 | 4 (20.0%)<br>20 | 4 (20.0%)<br>20 | 6 (30.0%)<br>20 | 3 (15.0%)<br>20 | 1 ( 5.0%)<br>20 | 0 ( 0.0%)<br>20 | 32 (20.0%)<br>160 |
| | Haemolysis<br>- Visual | | | | | | | | | |
| | (Yes/No)<br>No | 6 (30.0%) | 10 (50.0%) | 15 (75.0%) | 11 (55.0%) | 12 (60.0%) | 13 (65.0%) | 19 (95.0%) | 20 (100.0%) | 106 (66.2%) |
| | Yes<br>Total | 14 (70.0%)<br>20 | 10 (50.0%) | 5 (25.0%)<br>20 | 9 (45.0%) | 8 (40.0%)<br>20 | 7 (35.0%) | 1 (5.0%) | 0 ( 0.0%) | 54 (33.8%) |
| 6 | cfHb (mg/dL) | | | | | | | | - | |
| | Mean<br>95% Mean<br>CI | $191.24 \\171.53, 208.22$ | $188.75 \\ 165.51, 209.21$ | $166.15 \\ 150.82, 181.25$ | $172.37 \\158.32, 186.25$ | $173.04 \\ 159.51, 189.07$ | 170.39<br>155.95, 184.03 | $145.77 \\ 137.91, 153.45$ | $152.51 \\ 141.88, 162.78$ | $169.50 \\ 163.72, 175.30$ |
| | Median | 188.49 | 199.50 | 168.11 | 164.19 | 163.48 | 176.50 | 145.60 | 153.00 | 165.28 |
| | SD | 41.29 | 48.75 | 35.17 | 31.34 | 35.02 | 32.98 | 17.97 | 24.42 | 36.51 |
| | Min, Max<br>Total<br>Count | 75.26, 250.08<br>18 | 64.44, 276.65<br>18 | 96.55, 218.81<br>19 | 108.5, 221.35<br>18 | 119.11, 280.54<br>20 | 98.34, 215.76<br>20 | 115.71, 179.55<br>20 | 101.31, 205.98<br>20 | 64.44, 280.54<br>153 |
| | Haemolysis | | | | | | | | | |
| | - AU480<br>(Yes/No) | | | | | | | | | |
| | No | 11 (61.1%) | 9 (50.0%) | 16 (84.2%) | 13 (72.2%) | 17 (85.0%) | 16 (80.0%) | 20 (100.0%) | 19 (95.0%) | 121 (79.1%) |
| | Yes<br>Total | 7 (38.9%)<br>18 | 9 (50.0%)<br>18 | 3 (15.8%)<br>19 | 5 (27.8%)<br>18 | 3 (15.0%)<br>20 | 4 (20.0%)<br>20 | 0 ( 0.0%)<br>20 | 1 ( 5.0%)<br>20 | 32 (20.9%)<br>153 |
| | Haemolysis<br>- Visual | | | | | | | | | |
| | (Yes/No)<br>No | 6 (33.3%) | 5 (27.8%) | 12 (63.2%) | 11 (61.1%) | 13 (65.0%) | 10 (50.0%) | 20 (100.0%) | 18 (90.0%) | 95 (62.1%) |
| | Yes | 12 (66.7%) | 13 (72.2%) | 7 (36.8%) | 7 (38.9%) | 7 (35.0%) | 10 (50.0%) | 0 ( 0.0%) | 2 (10.0%) | 58 (37.9%) |
| 0.4 | Total | 18 | 18 | 19 | 18 | 20 | 20 | 20 | 20 | 153 |
| 24 | cfHb (mg/dL)<br>Mean | 167.54 | 189.19 | 171.23 | 171.64 | 152.95 | 163.34 | 143.22 | 155.87 | 163.37 |
| | 95% Mean<br>CI | 143.70, 191.58 | 165.61, 213.07 | 161.63, 180.64 | 156.24, 187.69 | 131.63, 175.36 | 147.13, 180.21 | 134.65, 151.83 | 145.77, 165.09 | 157.14, 169.70 |
| | Median | 160.38 | 182.91 | 170.18 | 163.25 | 136.96 | 158.61 | 143.07 | 161.72 | 161.40 |
| | SD<br>Min, Max | 50.25<br>68.3, 248.91 | 50.21<br>116.04, 283.39 | 21.05 $128.92, 208.47$ | $\begin{array}{c} 34.06 \\ 116.1,\ 232.11 \end{array}$ | 51.48<br>59.98, 271.69 | 38.17<br>84.58, 243.42 | 20.33<br>106.41, 179.48 | 22.85<br>106.81, 182.01 | 39.02<br>59.98, 283.39 |
| | Total<br>Count | 16 | 16 | 18 | 17 | 20 | 19 | 20 | 20 | 146 |
| | Haemolysis<br>- AU480 | | | | | | | | | |
| | (Yes/No)<br>No | 12 (75.0%) | 10 (62.5%) | 16 (88.9%) | 13 (76.5%) | 15 (75.0%) | 16 (84.2%) | 20 (100.0%) | 20 (100.0%) | 32 (83 60%) |
| | Yes | 4 (25.0%) | 6 (37.5%) | 2 (11.1%) | 4 (23.5%) | 5 (25.0%) | 3 (15.8%) | 0 ( 0.0%) | 0 ( 0.0%) | 24 (16.4%) |
| | Total | 16 | 16 | 18 | 17 | 20 | 19 | 20 | 20 | 146 |

Table A.8.1: Numerical Summary of Subjects Blood Analysis, for each time point, per Device Configuration (Gauge and Length) and Vacutainer tube and Overall continued

| Time<br>Point<br>(hours) | Characteristic | BD Nexiva (22G<br>x 1 inch) - 2mL | BD Nexiva (22G<br>x 1 inch) - 6mL | BD Nexiva (22G<br>x 1.75 inch) -<br>2mL | BD Nexiva (22G<br>x 1.75 inch) -<br>6mL | BD Nexiva (20G<br>x 1 inch) - 2mL | BD Nexiva (20G<br>x 1 inch) - 6mL | BD Nexiva (20G<br>x 1.75 inch) -<br>2mL | BD Nexiva (20G<br>x 1.75 inch) -<br>6mL | Overal |
|---|---|---|---|---|---|---|---|---|---|---|
| nours | Haemolysis - Visual | | | 211112 | OHL | | | 211111 | OHIL | |
| | (Yes/No) | | | | | | | | | |
| | No<br>Yes | 10 (62.5%)<br>6 (37.5%) | 8 (50.0%)<br>8 (50.0%) | 12 (66.7%)<br>6 (33.3%) | 11 (64.7%)<br>6 (35.3%) | 15 (75.0%)<br>5 (25.0%) | 14 (73.7%)<br>5 (26.3%) | 20 (100.0%)<br>0 ( 0.0%) | 18 (90.0%)<br>2 (10.0%) | 108 (74.0%<br>38 (26.0% |
| | Yes | 6 (37.5%) | 8 (50.0%) | 6 (33.3%) | 6 (35.3%) | 5 (25.0%) | 5 (26.3%) | 0 ( 0.0%) | 2 (10.0%) | 38 (26.0%) |
| 20 | Total<br>cfHb (mg/dL) | 16 | 16 | 18 | 17 | 20 | 19 | 20 | 20 | 140 |
| 30 | Mean | 185.52 | 210.60 | 167.79 | 169.92 | 158.51 | 162.12 | 153.68 | 150.67 | 166.8 |
| | 95% Mean | 156.51, 212.85 | 184.63, 239.48 | 151.42, 183.66 | 158.34, 182.34 | 140.63, 177.80 | 145.08, 178.00 | 146.47, 161.67 | 141.87, 159.93 | 160.26, 173.3 |
| | CI | 100.01, 212.00 | 101100, 200110 | 101.12, 100.00 | 100101, 102101 | 110.00, 111.00 | 110.00, 110.00 | 110:11, 101:01 | 111.01, 100.00 | 100.20, 110.0 |
| | Median | 196.62 | 197.89 | 173.95 | 169.28 | 150.21 | 164.66 | 148.96 | 148.17 | 162.7 |
| | SD | 54.86 | 50.87 | 34.25 | 25.29 | 42.43 | 37.41 | 17.77 | 21.35 | 38.8 |
| | Min, Max<br>Total | 92.32, 255.62<br>13 | 132.23, 298.24<br>12 | 110.07, 213.18<br>16 | 133.8, 228.66<br>16 | 81.58, 247.7<br>19 | 69.02, 250.81<br>19 | 124.97, 200.12<br>20 | 123.78, 188.76<br>20 | 69.02, 298.2 |
| | Count | 13 | 12 | 10 | 10 | 19 | 19 | 20 | 20 | 13 |
| | Haemolysis | | | | | | | | | |
| | Haemolysis<br>- AU480 | | | | | | | | | |
| | (Yes/No) | | | | | | | | | |
| | No | 7 (53.8%) | 7 (58.3%)<br>5 (41.7%) | 12 (75.0%)<br>4 (25.0%) | 14 (87.5%)<br>2 (12.5%) | 16 (84.2%)<br>3 (15.8%) | 17 (89.5%)<br>2 (10.5%) | 19 (95.0%)<br>1 ( 5.0%) | 20 (100.0%)<br>0 ( 0.0%) | 112 (83.0%<br>23 (17.0% |
| | $_{ m Yes}$ $_{ m Total}$ | 6 (46.2%)<br>13 | 5 (41.7%)<br>12 | 4 (25.0%)<br>16 | 2 (12.5%)<br>16 | 3 (15.8%)<br>19 | 2 (10.5%)<br>19 | 1 ( 5.0%) | 0 ( 0.0%) | 23 (17.0%<br>13 |
| | Haomolyeis | 15 | 12 | 10 | 10 | 19 | 19 | 20 | 20 | 13 |
| | Haemolysis<br>- Visual | | | | | | | | | |
| | (Yes/No) | | | | | | | | | |
| | No | 6 (46.2%) | 3 (25.0%) | 10 (62.5%) | 11 (68.8%)<br>5 (31.2%) | 13 (68.4%) | 14 (73.7%) | 18 (90.0%) | 16 (80.0%) | 91 (67.4%<br>44 (32.6% |
| | Yes | 7 (53.8%) | 9 (75.0%) | 6 (37.5%) | 5 (31.2%) | 6 (31.6%) | 5 (26.3%) | 2 (10.0%) | 4 (20.0%) | 44 (32.6% |
| 48 | Total<br>cfHb (mg/dL) | 13 | 12 | 16 | 16 | 19 | 19 | 20 | 20 | 13 |
| 48 | Mean | 212.51 | 219.02 | 178.49 | 174.76 | 158.17 | 168.39 | 148.86 | 149.54 | 169.3 |
| | 95% Mean | 190.93, 234.07 | 195.34, 245.23 | 166.08, 190.73 | 158.24, 190.35 | 143.31, 173.95 | 152.88, 184.93 | 143.20, 154.62 | 142.42, 156.99 | 163.17, 175.7 |
| | CI | | | | | | | | , | |
| | Median | 215.34 | 209.73 | 180.08 | 175.33 | 151.59 | 167.16 | 149.97 | 146.95 | 161.69 |
| | SD<br>Min, Max | 34.84 | 38.74 | 25.15 | 32.48 | 32.70 | 33.84 | 13.33 | 17.01 | 34.7 |
| | Min, Max<br>Total | 157.99, 269.46<br>9 | 175.61, 284.53<br>8 | 135.55, 212.02<br>15 | 110.22, 233.24<br>15 | 94.86, 223.68<br>16 | 116.07, 242.81<br>16 | 129.66, 170.4<br>20 | 119.31, 188.16<br>20 | 94.86, 284.5<br>11 |
| | Count | 9 | 0 | 10 | 10 | 10 | 10 | 20 | 20 | - 11 |
| | Haemolysis | | | | | | | | | |
| | - AU480 | | | | | | | | | |
| | (Yes/No)<br>No | - / | - / | | | | | / | / | |
| | No<br>Yes | 2 (22.2%)<br>7 (77.8%) | 3 (37.5%)<br>5 (62.5%) | 10 (66.7%)<br>5 (33.3%) | 12 (80.0%)<br>3 (20.0%) | 14 (87.5%) 2 (12.5%) | 13 (81.2%)<br>3 (18.8%) | 20 (100.0%)<br>0 ( 0.0%) | 20 (100.0%)<br>0 ( 0.0%) | 94 (79.0%<br>25 (21.0% |
| | Total | 7 (77.8%) | 5 (62.5%)<br>8 | 5 (55.5%)<br>15 | 3 (20.0%)<br>15 | 2 (12.5%) | 3 (18.8%) | 20 | 20 | 25 (21.0%<br>11 |
| | Haemolysis | <u> </u> | | 10 | 10 | 10 | 10 | 20 | 20 | - 11 |
| | - Visual | | | | | | | | | |
| | (Yes/No) | | | | | | | | | |
| | No | 2 (22.2%) | 2 (25.0%) | 7 (46.7%) | 8 (53.3%)<br>7 (46.7%) | 13 (81.2%) | 11 (68.8%) | 20 (100.0%) | 19 (95.0%) | 82 (68.9% |
| | Yes<br>Total | 7 (77.8%) | 6 (75.0%)<br>8 | 8 (53.3%)<br>15 | 7 (46.7%)<br>15 | 3 (18.8%)<br>16 | 5 (31.2%)<br>16 | 0 ( 0.0%) | 1 (5.0%) | 37 (31.1%<br>11 |
| 54 | cfHb (mg/dL) | | | 10 | 10 | 10 | 10 | 20 | 20 | |
| 01 | Mean | 180.69 | 220.07 | 166.77 | 164.29 | 170.58 | 151.13 | 144.48 | 154.89 | 162.7 |
| | 95% Mean | 157.23, 208.83 | 186.70, 252.39 | 148.36, 184.87 | 149.35, 177.62 | 147.01, 194.87 | 132.11, 168.79 | 136.31, 152.67 | 146.58, 163.53 | 156.17, 169.7 |
| | CI | | | | | | | | | |
| | $egin{array}{l} egin{array}{l} egin{array}$ | 167.93 | 222.47 | 165.77 | 172.10 | 169.55 | 149.39 | 146.47 | 151.33 | 159.2<br>35.5 |
| | Min, Max | $ \begin{array}{c} 36.32 \\ 141.72, 243.15 \end{array} $ | 48.41<br>169.64, 268.91 | $\begin{array}{c} 36.08 \\ 104.92,\ 222.54 \end{array}$ | $ \begin{array}{c} 27.18\\ 116.32, 196.82 \end{array} $ | $45.87 \\ 108.07, 250.53$ | 33.97 $94.07, 197.64$ | 18.73<br>116.47, 178.69 | $18.62 \\123.45, 194.23$ | 35.5<br>94.07 268.0 |
| | Total | 141.72, 243.13 | 109.04, 208.91 | 104.92, 222.34 | 13 | 108.07, 250.55 | 12 | 110.47, 178.09 | 123.45, 194.25 | 94.07, 268.9<br>10 |
| | Count | | | | -0 | | | | 10 | |
| | Haemolysis<br>- AU480 | | | | | | | | | |
| | - AU480 | | | | | | | | | |
| | (Yes/No) | | 0 (*0 001) | 11 (50 004) | 19 (100 007) | 10 (70 004) | 10 (100 007) | 10 (100 004) | 10 (100 00%) | 00 (00 10 |
| | NT. | | | | | | | | | |
| | (Yes/No)<br>No<br>Yes | 4 (66.7%)<br>2 (33.3%) | 3 (50.0%)<br>3 (50.0%) | 11 (78.6%)<br>3 (21.4%) | 13 (100.0%)<br>0 ( 0.0%)<br>13 | 10 (76.9%)<br>3 (23.1%) | 12 (100.0%)<br>0 ( 0.0%) | 19 (100.0%)<br>0 ( 0.0%) | 18 (100.0%)<br>0 ( 0.0%) | 90 (89.1%<br>11 (10.9% |

Table A.8.1: Numerical Summary of Subjects Blood Analysis, for each time point, per Device Configuration (Gauge and Length) and Vacutainer tube and Overall continued

| Time<br>Point<br>(hours) | Characteristic | BD Nexiva (22G<br>x 1 inch) - 2mL | BD Nexiva (22G<br>x 1 inch) - 6mL | BD Nexiva (22G<br>x 1.75 inch) -<br>2mL | BD Nexiva (22G<br>x 1.75 inch) -<br>6mL | BD Nexiva (20G<br>x 1 inch) - 2mL | BD Nexiva (20G<br>x 1 inch) - 6mL | BD Nexiva (20G<br>x 1.75 inch) -<br>2mL | BD Nexiva (20G<br>x 1.75 inch) -<br>6mL | Overall |
|---|---|---|---|---|---|---|---|---|---|---|
| ( 1 1 1 1 ) | Haemolysis - Visual | | | | - | | | | | |
| | (Yes/No) | | | | | | | | | |
| | No | 4 (66.7%) | 2 (33.3%) | 8 (57.1%) | 8 (61.5%) | 7 (53.8%) | 9 (75.0%) | 19 (100.0%) | 16 (88.9%) | 73 (72.3%) |
| | Yes | 2 (33.3%) | 4 (66.7%) | 6 (42.9%) | 5 (38.5%) | 6 (46.2%) | 3 (25.0%) | 0 ( 0.0%) | 2 (11.1%) | 28 (27.7%) |
| | Total | 6 | 6 | 14 | 13 | 13 | 12 | 19 | 18 | 101 |
| 72 | cfHb (mg/dL) | | | | | | | | | |
| | Mean | 184.83 | 211.15 | 190.26 | 181.81 | 143.39 | 185.70 | 148.12 | 138.60 | 165.03 |
| | 95% Mean<br>CI | 156.46, 214.29 | 171.81, 250.48 | 175.38, 204.42 | 154.09, 209.57 | 129.77, 162.99 | 155.46, 213.94 | 136.82, 159.65 | 129.95, 147.59 | 156.23, 174.25 |
| | Median | 180.15 | 204.68 | 198.61 | 177.06 | 135.06 | 202.90 | 138.18 | 142.76 | 153.87 |
| | SD | 40.42 | 49.86 | 21.32 | 41.43 | 27.98 | 45.62 | 24.00 | 16.89 | 38.68 |
| | Min, Max | 134.72, 235.61 | 156.91, 270.1 | 158.71, 217.83 | 128.38, 236.34 | 120.09, 213 | 110.75, 239.34 | 122.85, 182.83 | 118.5, 168.81 | 110.75, 270.1 |
| | Total | 6 | 5 | 7 | 7 | 9 | 8 | 16 | 13 | 71 |
| | Count | | | | | | | | | |
| | Haemolysis<br>- AU480 | | | | | | | | | |
| | (Yes/No) | 4 (00 =07) | 0 (40 00%) | 4 (55 107) | 4 (55 104) | 0 (00 00) | 1 (50 00) | 10 (100 0%) | 10 (100 00%) | FF (FF F04) |
| | No<br>Yes | 4 (66.7%)<br>2 (33.3%) | 2 (40.0%)<br>3 (60.0%) | 4 (57.1%)<br>3 (42.9%) | 4 (57.1%)<br>3 (42.9%) | 8 (88.9%)<br>1 (11.1%) | 4 (50.0%)<br>4 (50.0%) | 16 (100.0%)<br>0 ( 0.0%) | 13 (100.0%)<br>0 ( 0.0%) | 55 (77.5%)<br>16 (22.5%) |
| | Total | 2 (33.3%) | 3 (60.0%) | 3 (42.9%) | 3 (42.9%) | 1 (11.170) | 4 (50.0%) | 16 | 0 ( 0.0%) | 71 |
| | Haemolysis | 0 | 3 | ' | ' | | 0 | 10 | 13 | 11 |
| | - Visual | | | | | | | | | |
| | (Yes/No) | | | | | | | | | |
| | No | 3 (50.0%) | 2 (40.0%) | 2 (28.6%) | 4 (57.1%) | 8 (88.9%) | 3 (37.5%) | 14 (87.5%) | 13 (100.0%) | 49 (69.0%) |
| | Yes | 3 (50.0%) | 3 (60.0%) | 5 (71.4%) | 3 (42.9%) | 1 (11.1%) | 5 (62.5%) | 2 (12.5%) | 0 (0.0%) | 22 (31.0%) |
| | Total | ` <u>´</u> | ` ź | ` | ` | ` ģ | ` <u></u> | 16 | 13 | ` 71 |



#### A.9 Blood Draw Fill Time

Table A.9.1: Numerical Summary of Blood Draw Fill Time in seconds for each Vacutainer tube, per Device Configuration (Gauge and Length) and Overall

| tube | Characteristic | BD Nexiva (22G x 1 inch) | BD Nexiva (22G x 1.75 inch) | BD Nexiva (20G x 1 inch) | BD Nexiva (20G x 1.75 inch) | Overall |
|---|---|---|---|---|---|---|
| 2mL | Blood Draw Fill Time (sec) | · | | | | |
| | Mean | 59.30 | 60.29 | 59.53 | 60.95 | 60.10 |
| | 95% Mean CI | 58.23, 60.33 | 59.36, 61.20 | 58.67, 60.39 | 60.06, 61.82 | 59.64, 60.57 |
| | Median | 59.27 | 60.16 | 59.37 | 61.52 | 60.00 |
| | $\operatorname{SD}$ | 5.08 | 4.91 | 4.82 | 5.25 | 5.05 |
| | Min, Max | 45.83, 72.19 | 46.29, 73.76 | 46.69, 70.86 | 48.88, 77.06 | 45.83, 77.06 |
| | Total Count | 88 | 109 | 117 | 135 | 449 |
| 6mL | Blood Draw Fill Time (sec) | | | | | |
| | Mean | 100.29 | 100.60 | 99.14 | 98.97 | 99.67 |
| | 95% Mean CI | 98.90, 101.73 | 99.15, 101.98 | 97.77, 100.49 | 97.83, 100.16 | 98.99, 100.33 |
| | Median | 99.29 | 101.14 | 99.48 | 97.99 | 99.33 |
| | $\operatorname{SD}$ | 6.74 | 7.44 | 7.37 | 6.90 | 7.14 |
| | Min, Max | 84.03, 118.89 | 82.55, 118.55 | 84.03, 115.48 | 84.56, 119.35 | 82.55, 119.35 |
| | Total Count | 85 | 106 | 114 | 131 | 436 |

Table A.9.2: Numerical Summary of Blood Draw Fill Time in seconds for each Vacutainer tube, for each time point, per Device Configuration (Gauge and Length) and Vacutainer tube and Overall

| Tube | Time Point (hours) | Characteristic | BD Nexiva (22G x 1 inch) | BD Nexiva (22G x 1.75 inch) | BD Nexiva (20G x 1 inch) | BD Nexiva (20G x 1.75 inch) | Overall |
|---|---|---|---|---|---|---|---|
| 2mL | 0 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 58.77 | 61.25 | 60.41 | 59.01 | 59.86 |
| | | 95% Mean CI | 57.34, 60.13 | 59.28, 63.32 | 58.37, 62.49 | 56.57, 61.52 | 58.83, 60.89 |
| | | Median | 58.92 | 61.46 | 60.54 | 58.64 | 59.34 |
| | | SD | 3.29 | 4.70 | 4.87 | 5.69 | 4.74 |
| | | Min, Max | 51.27, 63.83 | 53.66, 70.59 | 51.38, 69.45 | 49.33, 69.93 | 49.33, 70.59 |
| | | Total Count | 20 | 20 | 20 | 20 | 80 |
| 2mL | 6 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 60.94 | 58.40 | 58.76 | 62.05 | 60.04 |
| | | 95% Mean CI | 59.21, 62.74 | 56.21, 60.58 | 57.19, 60.43 | 59.89, 64.32 | 59.03, 61.09 |
| | | Median | 59.90 | 59.05 | 58.06 | 62.15 | 59.43 |
| | | SD | 3.98 | 4.94 | 3.79 | 5.22 | 4.70 |
| | | Min, Max | 53.83, 68.83 | 46.29, 69.44 | 52.58, 65.84 | 52.49, 75.85 | 46.29, 75.85 |
| | | Total Count | 18 | 19 | 20 | 20 | 77 |
| 2mL | 24 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 56.85 | 60.95 | 58.56 | 60.95 | 59.41 |
| | | 95% Mean CI | 54.47, 59.10 | 58.49, 63.48 | 57.07, 60.08 | 58.34, 63.31 | 58.23, 60.56 |
| | | Median | 58.67 | 61.31 | 58.66 | 62.31 | 59.64 |
| | | SD | 4.92 | 5.57 | 3.54 | 5.82 | 5.21 |
| | | Min, Max | 48.08, 64.9 | 52.09, 72.58 | 50.83, 66.75 | 48.88, 68.39 | 48.08, 72.58 |
| | | Total Count | 16 | 18 | 20 | 20 | 74 |
| 2mL | 30 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 61.60 | 59.05 | 59.24 | 60.83 | 60.12 |
| | | 95% Mean CI | 58.68, 64.23 | 57.27, 60.80 | 57.19, 61.40 | 58.69, 63.00 | 58.99, 61.22 |
| | | Median | 61.98 | 59.51 | 58.57 | 60.79 | 60.00 |
| | | SD | 5.35 | 3.74 | 4.81 | 5.12 | 4.79 |
| | | Min, Max | 48.68, 69.78 | 53.62, 65.95 | 49.69, 70.86 | 51.25, 70.69 | 48.68, 70.86 |
| | | Total Count | 13 | 16 | 19 | 20 | 68 |



Table A.9.2: Numerical Summary of Blood Draw Fill Time in seconds for each Vacutainer tube, for each time point, per Device Configuration (Gauge and Length) and Vacutainer tube and Overall continued

| Tube | Time Point (hours) | Characteristic | BD Nexiva (22G x 1 inch) | BD Nexiva (22G x 1.75 inch) | BD Nexiva (20G x 1 inch) | BD Nexiva (20G x 1.75 inch) | Overall |
|---|---|---|---|---|---|---|---|
| 2mL | 48 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 59.11 | 60.82 | 59.95 | 62.41 | 60.86 |
| | | 95% Mean CI | 54.40, 63.75 | 59.28, 62.22 | 56.89, 62.73 | 60.51, 64.39 | 59.48, 62.16 |
| | | Median | 59.57 | 61.03 | 60.23 | 61.85 | 60.73 |
| | | SD | 7.70 | 3.04 | 6.27 | 4.47 | 5.31 |
| | | Min, Max | 45.83, 72.19 | 54.24, 65.8 | 46.69, 67.65 | 55.83, 73.5 | 45.83, 73.5 |
| | | Total Count | 9 | 15 | 16 | 20 | 60 |
| nL | 54 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 57.51 | 60.69 | 59.66 | 60.80 | 60.11 |
| | | 95% Mean CI | 53.32, 61.67 | 57.75, 63.88 | 56.50, 62.79 | 58.77, 62.72 | 58.66, 61.60 |
| | | Median | 57.25 | 58.89 | 61.26 | 62.02 | 61.07 |
| | | SD | 5.84 | 6.02 | 5.97 | 4.59 | 5.43 |
| | | Min, Max | 49.39, 65.32 | 49.53, 73.76 | 49.17, 68.98 | 51.95, 68.15 | 49.17, 73.76 |
| | | Total Count | 6 | 14 | 13 | 19 | 52 |
| nL | 72 | Blood Draw Fill Time (sec) | 0 | 14 | 10 | 19 | 32 |
| ш | 12 | Mean Mean | 59.78 | 61.94 | 61.16 | 60.52 | 60.82 |
| | | 95% Mean CI | 55.13, 63.86 | 57.39, 66.20 | 57.83, 64.25 | 58.00, 63.49 | 59.04, 62.61 |
| | | Median | 60.20 | 61.65 | 62.14 | 61.05 | 61.56 |
| | | SD | 5.99 | 6.54 | 5.25 | 5.87 | 5.67 |
| | | Min, Max | 49.86, 66.61 | 51.2, 70 | 52.68, 67.56 | 53.7, 77.06 | 49.86, 77.06 |
| | | Total Count | 6 | 7 | 9 | 16 | 38 |
| ıL | 0 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 98.51 | 98.75 | 96.41 | 98.84 | 98.13 |
| | | 95% Mean CI | 95.59, 101.39 | 95.38, 102.18 | 93.48, 99.30 | 95.70, 101.94 | 96.55, 99.67 |
| | | Median | 98.97 | 96.66 | 97.19 | 97.70 | 98.08 |
| | | SD | 6.80 | 8.05 | 6.76 | 7.36 | 7.19 |
| | | Min, Max | 84.03, 112.86 | 82.55, 112.09 | 84.24, 110.49 | 84.56, 115.29 | 82.55, 115.29 |
| | | Total Count | 20 | 20 | 20 | 20 | 80 |
| ıL | 6 | Blood Draw Fill Time (sec) | 20 | 20 | 20 | 20 | 00 |
| LL | 6 | Mean Mean | 101.60 | 97.88 | 101.11 | 99.86 | 100.13 |
| | | 95% Mean CI | | | | | |
| | | | 98.10, 105.23 | 94.19, 101.56 | 97.86, 104.39 | 96.86, 102.68 | 98.43, 101.82 |
| | | Median | 99.10 | 99.15 | 102.04 | 99.57 | 99.61 |
| | | SD | 8.02 | 8.07 | 7.64 | 6.77 | 7.60 |
| | | Min, Max | 84.14, 115.25 | 85.32, 111.59 | 88.65, 114.36 | 85.37, 113.48 | 84.14, 115.25 |
| | | Total Count | 18 | 18 | 20 | 20 | 76 |
| ıL | 24 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 100.36 | 99.57 | 98.44 | 99.57 | 99.45 |
| | | 95% Mean CI | 98.03, 102.98 | 96.38, 103.02 | 95.35, 101.50 | 98.15, 101.16 | 98.16, 100.79 |
| | | Median | 99.59 | 99.91 | 100.11 | 98.67 | 99.58 |
| | | SD | 5.19 | 7.03 | 6.89 | 3.54 | 5.72 |
| | | Min, Max | 93.63, 112.08 | 89.85, 116.46 | 86.57, 111.26 | 95.3, 108.19 | 86.57, 116.46 |
| | | Total Count | 16 | 17 | 19 | 20 | 72 |
| ıL | 30 | Blood Draw Fill Time (sec) | | | | | . <del>-</del> |
| | 00 | Mean Mean | 102.86 | 103.11 | 100.07 | 97.88 | 100.64 |
| | | 95% Mean CI | 99.28, 106.87 | 101.19, 104.96 | 95.85, 104.16 | 94.85, 101.24 | 98.86, 102.4 |
| | | Median | 103.15 | 103.39 | 99.95 | 94.68 | 101.98 |
| | | SD | 7.06 | 3.96 | 9.59 | 7.48 | 7.60 |
| | | Min, Max | 92.33, 118.89 | 96.36, 109.89 | 84.03, 115.48 | 89.66, 116.71 | 84.03, 118.89 |
| - | | Total Count | 12 | 16 | 19 | 20 | 67 |
| пL | 48 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 99.82 | 102.54 | 100.42 | 100.89 | 101.04 |
| | | 95% Mean CI | 96.37, 103.42 | 98.47, 106.69 | 96.88, 103.91 | 97.84, 103.92 | 99.21, 102.87 |
| | | Median | 99.01 | 103.16 | 99.16 | 99.86 | 99.71 |
| | | SD | 5.52 | 8.37 | 7.45 | 7.13 | 7.25 |
| | | Min, Max | 92.46, 108.6 | 85.27, 118.55 | 87.77, 113.06 | 87.61, 111.31 | 85.27, 118.55 |
| | | Total Count | 8 | 15 | 16 | 20 | 59 |
| ıL | 54 | Blood Draw Fill Time (sec) | | | | | |
| _ | | Mean (Sec) | 101.97 | 102.69 | 99.12 | 98.57 | 100.21 |
| | | 95% Mean CI | 96.33, 107.41 | 99.67, 105.60 | 97.09, 101.31 | 94.83, 102.79 | 98.28, 102.10 |
| | | Median | 104.34 | 102.21 | 98.58 | 97.15 | 100.00 |
| | | SD | | | | | |
| | | | 7.89 | 5.72 | 3.87 | 8.77 | 6.98 |
| | | Min, Max<br>Total Count | 92.02, 112.6<br>6 | 91.76, 112.19 | 93.56, 107.26 | 85.32, 119.35 | 85.32, 119.35 |
| | | | | 13 | 12 | 18 | 49 |



Table A.9.2: Numerical Summary of Blood Draw Fill Time in seconds for each Vacutainer tube, for each time point, per Device Configuration (Gauge and Length) and Vacutainer tube and Overall continued

| Tube | Time Point (hours) | Characteristic | BD Nexiva (22G x 1 inch) | BD Nexiva (22G x 1.75 inch) | BD Nexiva (20G x 1 inch) | BD Nexiva (20G x 1.75 inch) | Overall |
|---|---|---|---|---|---|---|---|
| 6mL | 72 | Blood Draw Fill Time (sec) | | | | | |
| | | Mean | 95.07 | 101.64 | 97.92 | 96.13 | 97.57 |
| | | 95% Mean CI | 92.50, 97.64 | 94.92, 108.95 | 93.41, 102.73 | 92.96, 99.59 | 95.19, 100.10 |
| | | Median | 94.85 | 104.38 | 97.71 | 95.10 | 95.91 |
| | | SD | 3.29 | 10.30 | 7.11 | 6.43 | 7.30 |
| | | Min, Max | 91.29, 99.09 | 90.24, 118.23 | 88.42, 109.56 | 87.75, 109.13 | 87.75, 118.23 |
| | | Total Count | 5 | 7 | 8 | 13 | 33 |





Table A.9.3: ANOVA table for Blood Draw Duration linear mixed effect model

| | Chisq | Df | Pr(>Chisq) | Result |
|-----------------------|---------|-------|------------|-------------|
| (Intercept) | 1829.42 | 1.00 | < 0.001 | Significant |
| timepoint | 6.47 | 6.00 | 0.372 | NS |
| device | 2.21 | 3.00 | 0.53 | NS |
| tube | 420.57 | 1.00 | < 0.001 | Significant |
| timepoint:device | 14.15 | 18.00 | 0.719 | NS |
| timepoint:tube | 5.09 | 6.00 | 0.532 | NS |
| device:tube | 2.76 | 3.00 | 0.43 | NS |
| timepoint:device:tube | 13.80 | 18.00 | 0.742 | NS |

Table A.9.4: Multiple Comparisons Based on linear mixed effect model for Blood Draw Duration. Sidak's adjustement for multiple comparisons was used.

| Tube | Time (hours) | Contrast | Estimate | Lwr | Upr | p-value | Result |
|---|---|---|---|---|---|---|---|
| 2mL | 0 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -2.48 | -7.47 | 2.51 | 0.576 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | -1.64 | -6.64 | 3.36 | 0.834 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -0.24 | -5.24 | 4.76 | 0.999 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 0.84 | -4.16 | 5.84 | 0.973 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | 2.24 | -2.76 | 7.24 | 0.655 | NS |
| | | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 1.40 | -3.59 | 6.39 | 0.888 | NS |
| | 6 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | 2.55 | -2.64 | 7.75 | 0.585 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | 2.19 | -2.95 | 7.33 | 0.691 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -1.10 | -6.24 | 4.04 | 0.946 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | -0.36 | -5.43 | 4.71 | 0.998 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | -3.65 | -8.72 | 1.42 | 0.248 | NS |
| | | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -3.29 | -8.28 | 1.70 | 0.325 | NS |
| | 24 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -4.12 | -9.54 | 1.30 | 0.206 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | -1.73 | -7.03 | 3.58 | 0.836 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -4.12 | -9.43 | 1.19 | 0.189 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 2.39 | -2.75 | 7.53 | 0.628 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | -0.00 | -5.14 | 5.14 | 1 | NS |
| | | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -2.39 | -7.38 | 2.60 | 0.605 | NS |
| | 30 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | 2.54 | -3.35 | 8.43 | 0.683 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | 2.35 | -3.34 | 8.04 | 0.711 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 0.76 | -4.87 | 6.39 | 0.985 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | -0.19 | -5.55 | 5.18 | 1 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | -1.78 | -7.08 | 3.52 | 0.824 | NS |
| | | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -1.59 | -6.64 | 3.46 | 0.849 | NS |
| | 48 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -1.75 | -8.39 | 4.89 | 0.905 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | -0.86 | -7.44 | 5.71 | 0.987 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -3.33 | -9.67 | 3.00 | 0.528 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 0.89 | -4.79 | 6.56 | 0.978 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | -1.58 | -6.98 | 3.81 | 0.873 | NS |
| | | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -2.47 | -7.75 | 2.81 | 0.624 | NS |
| | 54 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -3.25 | -10.93 | 4.43 | 0.695 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | -2.17 | -9.95 | 5.61 | 0.889 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -3.35 | -10.73 | 4.03 | 0.645 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 1.08 | -4.99 | 7.15 | 0.968 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | -0.10 | -5.66 | 5.45 | 1 | NS |
| | | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -1.18 | -6.85 | 4.48 | 0.949 | NS |
| | 72 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -2.24 | -11.01 | 6.53 | 0.913 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | -1.37 | -9.69 | 6.95 | 0.974 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -0.80 | -8.35 | 6.76 | 0.993 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 0.87 | -7.08 | 8.82 | 0.992 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | 1.44 | -5.71 | 8.59 | 0.954 | NS |
| | | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 0.57 | -5.99 | 7.14 | 0.996 | NS |
| 6mL | 0 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -0.24 | -5.23 | 4.75 | 0.999 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | 2.11 | -2.90 | 7.11 | 0.7 | NS |
| | | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -0.33 | -5.33 | 4.67 | 0.998 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 2.34 | -2.66 | 7.34 | 0.623 | NS |
| | | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | -0.09 | -5.10 | 4.91 | 1 | NS |



| | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -2.44 | -7.42 | 2.55 | 0.591 | NS |
|---|---|---|---|---|---|---|
| 6 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | 3.72 | -1.54 | 8.98 | 0.264 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | 0.49 | -4.65 | 5.63 | 0.995 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 1.75 | -3.39 | 6.89 | 0.818 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | -3.23 | -8.37 | 1.91 | 0.368 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | -1.98 | -7.12 | 3.16 | 0.755 | NS |
| | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 1.25 | -3.73 | 6.24 | 0.916 | NS |
| 24 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | 0.77 | -4.73 | 6.27 | 0.984 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | 1.90 | -3.47 | 7.27 | 0.799 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 0.77 | -4.54 | 6.08 | 0.982 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 1.13 | -4.16 | 6.41 | 0.947 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | -0.00 | -5.22 | 5.22 | 1 | NS |
| | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -1.13 | -6.18 | 3.93 | 0.94 | NS |
| 30 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -0.25 | -6.28 | 5.77 | 1 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | 2.79 | -3.04 | 8.62 | 0.607 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 4.98 | -0.79 | 10.75 | 0.118 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 3.04 | -2.32 | 8.41 | 0.462 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | 5.23 | -0.07 | 10.54 | 0.054 | NS |
| | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 2.19 | -2.86 | 7.24 | 0.679 | NS |
| 48 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -2.76 | -9.66 | 4.13 | 0.73 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | -0.63 | -7.46 | 6.20 | 0.995 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -1.11 | -7.71 | 5.50 | 0.973 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 2.13 | -3.54 | 7.81 | 0.766 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | 1.66 | -3.73 | 7.05 | 0.857 | NS |
| | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -0.48 | -5.76 | 4.80 | 0.996 | NS |
| 54 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -0.78 | -8.55 | 6.98 | 0.994 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | 2.87 | -5.01 | 10.75 | 0.784 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 3.35 | -4.08 | 10.78 | 0.651 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 3.65 | -2.66 | 9.96 | 0.443 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | 4.13 | -1.60 | 9.87 | 0.248 | NS |
| | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 0.48 | -5.38 | 6.35 | 0.997 | NS |
| 72 | BD Nexiva (22G x 1 inch) - BD Nexiva (22G x 1.75 inch) | -6.57 | -15.81 | 2.67 | 0.258 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1 inch) | -2.76 | -11.75 | 6.24 | 0.859 | NS |
| | BD Nexiva (22G x 1 inch) - BD Nexiva (20G x 1.75 inch) | -1.09 | -9.40 | 7.22 | 0.987 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1 inch) | 3.82 | -4.35 | 11.99 | 0.624 | NS |
| | BD Nexiva (22G x 1.75 inch) - BD Nexiva (20G x 1.75 inch) | 5.48 | -1.92 | 12.88 | 0.225 | NS |
| | BD Nexiva (20G x 1 inch) - BD Nexiva (20G x 1.75 inch) | 1.67 | -5.42 | 8.75 | 0.93 | NS |

### A.10 Thrombus Occurrence

Table A.10.1: Numerical Summary of Thrombus Occurrence, per Device Configuration (Gauge and Length) and Overall

| · · | · | / <b>1</b> | | 0 | O |
|---|---|---|---|---|---|
| Characteristic | BD Nexiva (22G | BD Nexiva (22G | BD Nexiva (20G | BD Nexiva (20G | Overall |
| | x 1 inch) | x 1.75 inch) | x 1 inch) | x 1.75 inch) | |
| Thrombus | | | | | |
| (Yes/No | | | | | |
| Yes | 62 (63.3%) | 72 (62.1%) | 99 (79.8%) | 68 (49.3%) | 301 (63.2%) |
| No | 36 (36.7%) | 44 (37.9%) | 25 (20.2%) | 70 (50.7%) | 175 (36.8%) |
| Total | 98 | 116 | 124 | 138 | 476 |

Table A.10.2: Numerical Summary of Thrombus Analysis, for each time point, per Device Configuration (Gauge and Length) and Overall

| Time Point<br>(hours) | Characteristic | BD Nexiva (22G<br>x 1 inch) | BD Nexiva (22G<br>x 1.75 inch) | BD Nexiva (20G<br>x 1 inch) | BD Nexiva (20G<br>x 1.75 inch) | Overall |
|---|---|---|---|---|---|---|
| 0 | Thrombus | , | , , , | , | , | |
| | (Yes/No | | | | | |
| | Yes | 14 (70.0%) | 13 (65.0%) | 16 (80.0%) | 10 (50.0%) | 53 (66.2%) |
| | No | 6 (30.0%) | 7 (35.0%) | 4 (20.0%) | 10 (50.0%) | 27 (33.8%) |
| | Total | 20 | 20 | 20 | 20 | 80 |
| 6 | Thrombus | | | | | |
| | (Yes/No | | | | | |
| | Yes | 14 (70.0%) | 12 (63.2%) | 16 (80.0%) | 10 (50.0%) | 52 (65.8% |
| | No | 6 (30.0%) | 7 (36.8%) | 4 (20.0%) | 10 (50.0%) | 27 (34.2% |
| | Total | 20 | 19 | 20 | 20 | 79 |
| 24 | Thrombus | | | | | |
| | (Yes/No | | | | | |
| | Yes | 12 (66.7%) | 11 (61.1%) | 16 (80.0%) | 10 (50.0%) | 49 (64.5% |
| | No | 6 (33.3%) | 7 (38.9%) | 4 (20.0%) | 10 (50.0%) | 27 (35.5% |
| | Total | 18 | 18 | 20 | 20 | 7 |
| 30 | Thrombus | | | | | |
| | (Yes/No | | | | | |
| | Yes | 10 (62.5%) | 11 (64.7%) | 15 (78.9%) | 10 (50.0%) | 46 (63.9% |
| | No | 6 (37.5%) | 6 (35.3%) | 4 (21.1%) | 10 (50.0%) | 26 (36.1% |
| | Total | 16 | 17 | 19 | 20 | 7 |
| 48 | Thrombus | | | | | |
| | (Yes/No | 0 (54 504) | 10 (00 800) | 1 × (00 004) | 40 (80 00) | 11 (00 10) |
| | Yes | 6 (54.5%) | 10 (62.5%) | 15 (83.3%) | 10 (50.0%) | 41 (63.1% |
| | No | 5 (45.5%) | 6 (37.5%) | 3 (16.7%) | 10 (50.0%) | 24 (36.9% |
| | Total | 11 | 16 | 18 | 20 | 6- |
| 54 | Thrombus | | | | | |
| | (Yes/No | 9 (40 00%) | 0 (55 104) | 19 (01 007) | 10 (50 007) | 24 (50 007 |
| | Yes<br>No | 3 (42.9%) | 8 (57.1%) | 13 (81.2%) | 10 (50.0%)<br>10 (50.0%) | 34 (59.6% |
| | | 4 (57.1%)<br>7 | 6 (42.9%)<br>14 | 3 (18.8%)<br>16 | 10 (50.0%) | 23 (40.4%<br>5 |
| 72 | Total Thrombus | | 14 | 10 | 20 | 9 |
| 12 | (Yes/No | | | | | |
| | (Yes/No<br>Yes | 3 (50.0%) | 7 (58.3%) | 8 (72.7%) | 8 (44.4%) | 26 (55.3% |
| | Yes<br>No | 3 (50.0%) | 5 (41.7%) | 3 (27.3%) | 8 (44.4%)<br>10 (55.6%) | 20 (55.3%) |
| | Total | 3 (50.0%)<br>6 | 3 (41.7%) | 3 (27.3%)<br>11 | 10 (55.6%) | 4 (44.776 |
| | Iotai | 0 | 12 | 11 | 16 | 4 |





# **B** Figures

#### **B.1** Survival

Figure B.1.1: Survival Curve for Indwell Time per Device Configuration. Color bands represent 95% Confidence Intervals





### **B.2** Indwell Time



Figure B.2.1: Boxplot for Indwell Time per Device Configuration



#### **B.3** Blood Analysis

#### **B.3.1** cfHb

Figure B.3.1: Boxplot for cfHb per Device Configuration for each Timepoint





BD Nexiva (20G x 1 inch) BD Nexiva (20G x 1.75 inch) S002 S003 S006 S007 S011 S002 S003 S006 S007 S011 250 200 200 175 150 150 125 100 100 50 S012 S013 S020 S012 S013 S015 S017 S020 S015 S017 250 175 200 150 150 cfHb (mg/dL) cfHb (mg/dL) 125 100 100 50 S022 S024 S025 S026 S029 S022 S024 S025 S026 S029 250 200 200 175 150 150 125 100 100 50 S030 S034 S036 S037 S038 S030 S034 S036 S037 S038 250 200 175 200 150 150 125 100 100 0 24 48 72 0 24 48 72 0 24 48 72 0 24 48 72 0 0 24 48 72 0 24 48 72 0 24 48 72 0 24 48 72 0 24 48 72 24 48 72 Tube Time (hours) Time (hours) 🕶 2mL BD Nexiva (22G x 1 inch) BD Nexiva (22G x 1.75 inch) 6mL S001 S004 S005 S008 S009 S001 S004 S005 S008 S009 300 250 200 200 150 150 100 100 S010 S014 S016 S018 S019 S010 S014 S016 S018 S019 300 250 200 200 150 150 cfHb (mg/dL) cfHb (mg/dL) 100 S023 S031 S021 S023 S028 S031 S021 S027 S028 S027 300 250 200 200 150 150 100 100 S032 S033 S035 S039 S040 S032 S033 S035 S039 S040 300 250 200 200 150 150 100 100 0 24 48 72 0 24 48 72 0 24 48 72 0 24 48 72 0 24 48 72 72 0 24 48 72 0 24 48 72 0 24 48 72 0 24 48 72 0 24 48 Time (hours) Time (hours)

Figure B.3.2: Lineplot for cfHb per subject and Device Configuration over time



#### **B.4** Haemolysis Occurrence

Figure B.4.1: Barplot for Haemolysis Occurence (assessed with AU480) per Device Configuration





Figure B.4.2: Barplot for Haemolysis Occurence (AU480 measurements) per Device Configuration for each Timepoint





#### **B.5** Blood Draw Fill Time



Figure B.5.1: Boxplot for Blood Draw Fill Time per Device Configuration



Figure B.5.2: Estimated Blood Draw Fill Time Difference (with 95% CI) between Device Configurations for 2 and 6mL Vacutainer tubes





Figure B.5.3: Lineplot for Blood Draw Fill Time per Device Configuration at each captured timepoint



Figure B.5.4: Estimated Blood Draw Fill Time Difference (with 95% CI) between Device Configurations for 2 and 6mL Vacutainer tubes per Time Point







### **B.6** Thrombus Occurrence

Device

Figure B.6.1: Barplot for Thrombus Occurence per Device Configuration



BD Nexiva (22G x 1 inch) BD Nexiva (22G x 1.75 inch) 75% 50% Percentage of Thrombus (%) 0% 0% 75% BD Nexiva (20G x 1 inch) BD Nexiva (20G x 1.75 inch) 50% 25% 8 30 -8⁄2 6 \$ -8% 54 54 , N V Time (hours)

Figure B.6.2: Barplot for Thrombus Occurence per Device Configuration for each Timepoint



#### B.7 Feature Importance with Boruta Algorithm

Figure B.7.1: Boruta plot showing survival predictive importance of features

## Importance values for 80 observations



Note: The output of the Boruta algorithm represents the predictive importance of each feature. The algorithm statistically compares the importance of each feature to the importance of random features called "shadow variables" (obtained from the random permutation of the features available in the dataset). Features are assessed as being "Confirmed" when showing a significantly higher importance than the best shadow variables (shadowMax). For more details, please refer to [2].



device

adowMax

adowMax

adowMean

bength
hadowMin

bength
hadowMin

shadowMin

shadowMin

shadowMin

shadowMin

Figure B.7.2: Boruta plot showing evolution of predictive importance of features over time

Note: The output presented in Figure B.7.2 represents the evolution of the output of the Boruta algorithm when considering median importance of predictors for device failure observed up to any considered time point, therefore potentially showing how different predictors can predominantly be associated with failures over time.



# C Listings

Table C.0.1: Dummy randomization list (rows 1 to 40)

| | | one C.u. | | mmy random | nzauton | , | |
|---|---|---|---|---|---|---|---|
| subjID | randoID | gauge | order | arm_length | arm | length | device |
| S001 | 101001.00 | 22G | 1 | RA_1.75 inch | Right | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S001 | 101001.00 | 22G | 2 | $LA_{-1}$ inch | Left | 1 inch | BD Nexiva (22G x 1 inch) |
| S002 | 101002.00 | 20G | 1 | $LA_{-1.75}$ inch | Left | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S002 | 101002.00 | 20G | 2 | $RA_1$ inch | Right | 1 inch | BD Nexiva (20G x 1 inch) |
| S003 | 101003.00 | 20G | 1 | $LA_1$ inch | Left | 1 inch | BD Nexiva (20G x 1 inch) |
| S003 | 101003.00 | 20G | 2 | $RA_1.75$ inch | Right | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S004 | 101004.00 | 22G | 1 | $LA_{-1}$ inch | Left | 1 inch | BD Nexiva (22G x 1 inch) |
| S004 | 101004.00 | 22G | 2 | $RA_1.75$ inch | Right | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S005 | 101005.00 | 22G | 1 | RA_1 inch | Right | 1 inch | BD Nexiva (22G x 1 inch) |
| S005 | 101005.00 | 22G | 2 | $LA_1.75$ inch | Left | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S006 | 101006.00 | 20G | 1 | $RA_{-1.75}$ inch | Right | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S006 | 101006.00 | 20G | 2 | $LA_1$ inch | Left | 1 inch | BD Nexiva (20G x 1 inch) |
| S007 | 101007.00 | 20G | 1 | RA_1 inch | Right | 1 inch | BD Nexiva (20G x 1 inch) |
| S007 | 101007.00 | 20G | 2 | $LA_1.75$ inch | Left | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S008 | 101008.00 | 22G | 1 | $LA_{-1.75}$ inch | Left | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S008 | 101008.00 | 22G | 2 | $RA_1$ inch | Right | 1 inch | BD Nexiva (22G x 1 inch) |
| S009 | 101009.00 | 22G | 1 | $RA_1.75$ inch | Right | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S009 | 101009.00 | 22G | 2 | $LA_1$ inch | Left | 1 inch | BD Nexiva (22G x 1 inch) |
| S010 | 101010.00 | 22G | 1 | $LA_{-1}$ inch | Left | 1 inch | BD Nexiva (22G x 1 inch) |
| S010 | 101010.00 | 22G | 2 | $RA_1.75$ inch | Right | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S011 | 101011.00 | 20G | 1 | $RA_1$ inch | Right | 1 inch | BD Nexiva (20G x 1 inch) |
| S011 | 101011.00 | 20G | 2 | $LA_{-1.75}$ inch | Left | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S012 | 101012.00 | 20G | 1 | $LA_{-1}$ inch | Left | 1 inch | BD Nexiva (20G x 1 inch) |
| S012 | 101012.00 | 20G | 2 | $RA_1.75$ inch | Right | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S013 | 101013.00 | 20G | 1 | $RA_1.75$ inch | Right | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S013 | 101013.00 | 20G | 2 | $LA_1$ inch | Left | 1 inch | BD Nexiva (20G x 1 inch) |
| S014 | 101014.00 | 22G | 1 | $LA_1.75$ inch | Left | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S014 | 101014.00 | 22G | 2 | RA_1 inch | Right | 1 inch | BD Nexiva (22G x 1 inch) |
| S015 | 101015.00 | 20G | 1 | $LA_{-1.75}$ inch | Left | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S015 | 101015.00 | 20G | 2 | RA_1 inch | Right | 1 inch | BD Nexiva (20G x 1 inch) |
| S016 | 101016.00 | 22G | 1 | RA_1 inch | Right | 1 inch | BD Nexiva (22G x 1 inch) |
| S016 | 101016.00 | 22G | 2 | $LA_{-1.75}$ inch | Left | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S017 | 101017.00 | 20G | 1 | RA_1 inch | Right | 1 inch | BD Nexiva (20G x 1 inch) |
| S017 | 101017.00 | 20G | 2 | $LA_{-1.75}$ inch | Left | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S018 | 101018.00 | 22G | 1 | LA_1 inch | Left | 1 inch | BD Nexiva (22G x 1 inch) |
| S018 | 101018.00 | 22G | 2 | $RA_1.75$ inch | Right | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S019 | 101019.00 | 22G | 1 | $RA_1.75$ inch | Right | 1.75 inch | BD Nexiva (22G x 1.75 inch) |
| S019 | 101019.00 | 22G | 2 | LA_1 inch | Left | 1 inch | BD Nexiva (22G x 1 inch) |
| S020 | 101020.00 | 20G | 1 | $LA_1.75$ inch | Left | 1.75 inch | BD Nexiva (20G x 1.75 inch) |
| S020 | 101020.00 | 20G | 2 | RA_1 inch | Right | 1 inch | BD Nexiva (20G x 1 inch) |



Table C.0.2: Dummy Demographics listing (rows 1 to 40).

| Subjil S | 1.175 | | | | Jumny Demograpine | - \ | | . 1 . | |
|---|---|---|---|---|---|---|---|---|---|
| S002 20G 47,90 F Hispanic / Latino White / Caucasian 151,20 57,90 20,00 S003 20G 47,20 M Non Hispanic / Latino Other 159,00 59,00 19,00 S005 22G 57,10 F Non Hispanic / Latino Asian 165,20 68,10 20,00 S006 22G 57,10 F Non Hispanic / Latino Other 159,30 58,80 18,00 S007 20G 31,70 F Non Hispanic / Latino Asian 158,20 80,50 24,00 S008 22G 57,40 F Non Hispanic / Latino Other Caucasian 172,50 63,50 22,00 S010 22G 39,80 M Non Hispanic / Latino Other 174,40 65,50 25,00 S011 20G 54,40 F Non Hispanic / Latino Other 170,40 56,20 23,00 S013 20G 39,0 M Non Hispanic / L | | | | - | v | | - | | |
| Sond 20G | | | | | | | | | |
| Soul | | | | | | / | | | |
| S005 22G 57.10 F Non Hispanic / Latino White / Caucasian 160.30 76.30 20.00 | | | | | - , | | | | |
| S006 20G 56.30 F Non Hispanic / Latino Other 159.30 58.80 18.00 S007 20G 31.70 F Non Hispanic / Latino Asian Asian 172.50 63.50 22.00 S009 22G 32.90 F Non Hispanic / Latino Other 174.90 86.20 224.00 S010 22G 39.80 M Non Hispanic / Latino Asian 174.80 65.50 25.00 S011 20G 25.20 M Non Hispanic / Latino Asian 174.80 65.50 25.00 S012 20G 54.40 F Non Hispanic / Latino Other 170.40 56.20 23.00 S013 20G 43.40 F Non Hispanic / Latino Asian 177.10 74.20 23.00 S013 20G 43.40 F Non Hispanic / Latino Asian 177.10 74.20 23.00 S014 22G 28.50 M Non Hispanic / Latino Other 185.60 77.30 27.00 S015 20G 39.20 M Non Hispanic / Latino Other 185.60 77.30 27.00 S016 22G 32.50 F Non Hispanic / Latino Asian 150.40 69.10 24.00 S017 20G 25.40 F Non Hispanic / Latino Other 180.70 75.50 19.00 S018 22G 24.30 M Non Hispanic / Latino Other 180.70 75.50 19.00 S019 22G 25.50 M Non Hispanic / Latino Other 180.70 75.50 19.00 S019 22G 26.40 F Non Hispanic / Latino Asian 181.20 71.50 25.00 S018 22G 24.30 M Non Hispanic / Latino Asian 188.60 84.40 24.00 S020 20G 49.00 M Non Hispanic / Latino Asian 188.60 84.40 24.00 S020 20G 49.00 M Non Hispanic / Latino Asian 188.60 84.40 24.00 S022 20G 26.50 M Non Hispanic / Latino Asian 185.50 54.20 23.00 S023 22G 24.60 M Non Hispanic / Latino Asian 185.50 54.20 23.00 S023 22G 24.60 M Non Hispanic / Latino Asian 185.20 59.50 19.00 S026 22G 28.10 M Non Hispanic / Latino Asian 185.20 59.50 19.00 S026 22G 28.10 M Non Hispanic / Latino Other 156.30 79.90 23.00 S026 22G 26.50 M Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 26.50 M Non Hispanic / Latino Other 156.60 6 | | | | | | | | | |
| Sour | | | | | | , | | | |
| Source | | | | | | | | | |
| S009 22G 32.90 F Non Hispanic / Latino Asian 174.80 65.50 25.00 | | | | | | | | | |
| S010 22G 39.80 M Non Hispanic / Latino Asian 174.80 65.50 25.00 S011 20G 25.20 M Non Hispanic / Latino White / Caucasian 160.40 52.80 19.00 S012 20G 54.40 F Non Hispanic / Latino Asian 177.10 74.20 23.00 S014 22G 28.50 M Non Hispanic / Latino Asian 177.10 74.20 23.00 S015 20G 39.20 M Non Hispanic / Latino Other 185.60 77.30 27.00 S015 20G 39.20 M Non Hispanic / Latino Asian 155.50 73.70 26.00 S016 22G 25.40 F Non Hispanic / Latino White / Caucasian 181.20 71.50 25.00 S018 22G 24.30 M Non Hispanic / Latino White / Caucasian 181.20 71.50 25.00 S018 22G 24.30 M Non Hispanic / Latino White / Caucasian 180.70 75.50 19.00 S019 22G 55.50 M Non Hispanic / Latino White / Caucasian 183.60 84.40 24.00 S020 20G 49.00 M Non Hispanic / Latino White / Caucasian 153.50 54.20 23.00 S021 22G 28.30 M Non Hispanic / Latino White / Caucasian 153.50 54.20 23.00 S022 20G 46.00 F Non Hispanic / Latino Asian 184.50 76.80 20.00 S023 22G 54.60 M Non Hispanic / Latino Asian 184.50 76.80 20.00 S024 20G 24.20 M Non Hispanic / Latino S024 20G 24.20 M Non Hispanic / Latino S025 20G 28.10 M Non Hispanic / Latino Other 155.30 82.40 26.00 S025 20G 28.10 M Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino Other 152.50 77.70 25.00 S031 22G 26.50 M Non Hispanic / Latino Other 152.50 77.70 25.00 S032 22G 45.00 M Non Hispanic / Latino Other 152.50 77.70 25.00 S033 22G 25.50 M Non Hispanic / Latino Other 153.50 61.10 21.00 S036 20G 52.20 F Non Hispanic / Latino Other 153.50 61.10 21.00 S036 20G 29.90 F Hispanic / Latino Other 153.5 | | | | | - , | , | | | |
| S011 20G 25.20 M | | | | | - , | | | | |
| S012 20G 54.40 F Non Hispanic / Latino Other 170.40 56.20 23.00 S013 20G 43.40 F Non Hispanic / Latino Asian 177.10 74.20 23.00 S014 22G 28.50 M Non Hispanic / Latino White / Caucasian 155.50 73.70 26.00 S015 20G 39.20 M Non Hispanic / Latino Other 185.60 77.30 27.00 S016 22G 32.50 F Non Hispanic / Latino Other 180.40 69.10 24.00 S017 20G 25.40 F Non Hispanic / Latino Other 180.70 75.50 19.00 S018 22G 24.30 M Non Hispanic / Latino Other 180.70 75.50 19.00 S012 22G 25.50 M Non Hispanic / Latino Other 169.70 71.80 23.00 S021 22G 28.30 M Non Hispanic / Latino <td< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></td<> | | | | | | | | | |
| S013 20G 43.40 F Non Hispanic / Latino Asian 177.10 74.20 23.00 S014 22G 28.50 M Non Hispanic / Latino White / Caucasian 155.50 73.70 26.00 S015 20G 39.20 M Non Hispanic / Latino Other 185.60 77.30 27.00 S016 22G 32.50 F Non Hispanic / Latino Other 185.60 77.30 25.00 S017 20G 25.40 F Non Hispanic / Latino Other 180.70 75.50 19.00 S018 22G 24.30 M Non Hispanic / Latino Other 180.70 75.50 19.00 S019 22G 55.50 M Non Hispanic / Latino White / Caucasian 181.20 71.50 25.00 S020 20G 49.00 M Non Hispanic / Latino White / Caucasian 185.30 82.40 24.00 S022 20G 46.00 F Non Hispanic / | | | | | - , | , | | | |
| S014 22G 28.50 M Non Hispanic / Latino White / Caucasian 155.50 73.70 26.00 S015 20G 39.20 M Non Hispanic / Latino Other 185.60 77.30 27.00 S016 22G 32.50 F Non Hispanic / Latino Asian 150.40 69.10 24.00 S017 20G 25.40 F Non Hispanic / Latino White / Caucasian 181.20 71.50 25.00 S018 22G 24.30 M Non Hispanic / Latino Other 180.70 75.50 19.00 S019 22G 55.50 M Non Hispanic / Latino Asian 188.60 84.40 24.00 S021 22G 28.30 M Non Hispanic / Latino White / Caucasian 185.50 76.80 23.00 S022 20G 46.00 F Non Hispanic / Latino White / Caucasian 185.30 82.40 26.00 S024 20G 24.20 M No | | | | | - , | | | | |
| S015 20G 39.20 M Non Hispanic / Latino Other 185.60 77.30 27.00 S016 22G 32.50 F Non Hispanic / Latino Asian 150.40 69.10 24.00 S017 20G 25.40 F Non Hispanic / Latino White / Caucasian 181.20 71.50 25.00 S018 22G 24.30 M Non Hispanic / Latino Other 180.70 75.50 19.00 S019 22G 55.50 M Non Hispanic / Latino Asian 188.60 84.40 24.00 S020 20G 49.00 M Non Hispanic / Latino Other 169.70 71.80 23.00 S021 22G 28.30 M Non Hispanic / Latino Other 169.70 71.80 23.00 S022 20G 46.00 F Non Hispanic / Latino Other 156.30 79.90 23.00 S024 20G 24.20 M Non Hispanic / Latino <td< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></td<> | | | | | | | | | |
| S016 22G 32.50 F Non Hispanic / Latino Asian 150.40 69.10 24.00 S017 20G 25.40 F Non Hispanic / Latino White / Caucasian 181.20 71.50 25.00 S018 22G 24.30 M Non Hispanic / Latino Other 180.70 75.50 19.00 S019 22G 55.50 M Non Hispanic / Latino Asian 188.60 84.40 24.00 S020 20G 49.00 M Non Hispanic / Latino Other 169.70 71.80 23.00 S021 22G 28.30 M Non Hispanic / Latino Other 169.70 71.80 23.00 S022 20G 46.00 F Non Hispanic / Latino Other 169.70 71.80 23.00 S023 22G 54.60 M Non Hispanic / Latino Other 156.30 79.90 23.00 S024 20G 24.20 M Non Hispanic / Latino <td< td=""><td></td><td></td><td></td><td></td><td></td><td>,</td><td></td><td></td><td></td></td<> | | | | | | , | | | |
| S017 20G 25.40 F Non Hispanic / Latino White / Caucasian 181.20 71.50 25.00 S018 22G 24.30 M Non Hispanic / Latino Other 180.70 75.50 19.00 S019 22G 55.50 M Non Hispanic / Latino Asian 188.60 84.40 24.00 S020 20G 49.00 M Non Hispanic / Latino Other 169.70 71.80 23.00 S021 22G 28.30 M Non Hispanic / Latino Other 169.70 71.80 23.00 S022 20G 46.00 F Non Hispanic / Latino Asian 184.50 76.80 20.00 S023 22G 54.60 M Non Hispanic / Latino Other 156.30 79.90 23.00 S024 20G 24.20 M Non Hispanic / Latino Other 156.30 79.90 23.00 S025 20G 28.10 M Non Hispanic / Latino <td< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></td<> | | | | | | | | | |
| S018 22G 24.30 M Non Hispanic / Latino Other 180.70 75.50 19.00 S019 22G 55.50 M Non Hispanic / Latino Asian 188.60 84.40 24.00 S020 20G 49.00 M Non Hispanic / Latino White / Caucasian 153.50 54.20 23.00 S021 22G 28.30 M Non Hispanic / Latino Other 169.70 71.80 23.00 S022 20G 46.00 F Non Hispanic / Latino Other 169.70 71.80 23.00 S022 20G 46.00 F Non Hispanic / Latino Other 185.30 82.40 26.00 S023 22G 54.60 M Non Hispanic / Latino Other 156.30 79.90 23.00 S025 20G 28.10 M Non Hispanic / Latino Other 157.00 75.30 26.00 S027 22G 29.30 F Non Hispanic / Latino <td< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></td<> | | | | | | | | | |
| S019 22G 55.50 M Non Hispanic / Latino Asian 188.60 84.40 24.00 S020 20G 49.00 M Non Hispanic / Latino White / Caucasian 153.50 54.20 23.00 S021 22G 28.30 M Non Hispanic / Latino Other 169.70 71.80 23.00 S022 20G 46.00 F Non Hispanic / Latino Asian 184.50 76.80 20.00 S023 22G 54.60 M Non Hispanic / Latino Other 156.30 79.90 23.00 S024 20G 24.20 M Non Hispanic / Latino Other 156.30 79.90 23.00 S025 20G 28.10 M Non Hispanic / Latino Asian 185.20 59.50 19.00 S026 20G 55.10 M Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino <td< td=""><td></td><td></td><td></td><td></td><td>- ,</td><td>,</td><td></td><td></td><td></td></td<> | | | | | - , | , | | | |
| S020 20G 49.00 M Non Hispanic / Latino White / Caucasian 153.50 54.20 23.00 S021 22G 28.30 M Non Hispanic / Latino Other 169.70 71.80 23.00 S022 20G 46.00 F Non Hispanic / Latino Asian 184.50 76.80 20.00 S023 22G 54.60 M Non Hispanic / Latino White / Caucasian 185.30 82.40 26.00 S024 20G 24.20 M Non Hispanic / Latino Other 156.30 79.90 23.00 S025 20G 28.10 M Non Hispanic / Latino Asian 185.20 59.50 19.00 S026 20G 55.10 M Non Hispanic / Latino Other 157.00 75.30 26.00 S027 22G 29.30 F Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino | | | | | | | | | |
| S021 22G 28.30 M Non Hispanic / Latino Other 169.70 71.80 23.00 S022 20G 46.00 F Non Hispanic / Latino Asian 184.50 76.80 20.00 S023 22G 54.60 M Non Hispanic / Latino White / Caucasian 185.30 82.40 26.00 S024 20G 24.20 M Non Hispanic / Latino Other 156.30 79.90 23.00 S025 20G 28.10 M Non Hispanic / Latino Asian 185.20 59.50 19.00 S026 20G 55.10 M Non Hispanic / Latino White / Caucasian 161.70 75.30 26.00 S027 22G 29.30 F Non Hispanic / Latino Asian 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino White / Caucasian 170.70 81.60 21.00 S030 20G 52.30 F Non Hispanic / | | | | | | | | | |
| S022 20G 46.00 F Non Hispanic / Latino Asian 184.50 76.80 20.00 S023 22G 54.60 M Non Hispanic / Latino White / Caucasian 185.30 82.40 26.00 S024 20G 24.20 M Non Hispanic / Latino Other 156.30 79.90 23.00 S025 20G 28.10 M Non Hispanic / Latino Asian 185.20 59.50 19.00 S026 20G 55.10 M Non Hispanic / Latino White / Caucasian 161.70 75.30 26.00 S027 22G 29.30 F Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino Asian 155.20 84.20 24.00 S030 20G 52.30 F Non Hispanic / Latino Other 152.50 77.70 25.00 S031 22G 26.50 M Non Hispanic / Latino | | | | | - , | , | | | |
| S023 22G 54.60 M Non Hispanic / Latino White / Caucasian 185.30 82.40 26.00 S024 20G 24.20 M Non Hispanic / Latino Other 156.30 79.90 23.00 S025 20G 28.10 M Non Hispanic / Latino Asian 185.20 59.50 19.00 S026 20G 55.10 M Non Hispanic / Latino White / Caucasian 161.70 75.30 26.00 S027 22G 29.30 F Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino Asian 155.20 84.20 24.00 S029 20G 44.30 M Non Hispanic / Latino White / Caucasian 170.70 81.60 21.00 S031 22G 26.50 M Non Hispanic / Latino Other 152.50 77.70 25.00 S032 22G 45.00 M Non Hispanic / | | | | | | | | | |
| S024 20G 24.20 M Non Hispanic / Latino Other 156.30 79.90 23.00 S025 20G 28.10 M Non Hispanic / Latino Asian 185.20 59.50 19.00 S026 20G 55.10 M Non Hispanic / Latino White / Caucasian 161.70 75.30 26.00 S027 22G 29.30 F Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino Asian 155.20 84.20 24.00 S029 20G 44.30 M Non Hispanic / Latino White / Caucasian 170.70 81.60 21.00 S030 20G 52.30 F Non Hispanic / Latino Other 152.50 77.70 25.00 S031 22G 26.50 M Non Hispanic / Latino Asian 178.80 69.60 25.00 S032 22G 45.00 M Non Hispanic / Latino | | | | | | | | | |
| S025 20G 28.10 M Non Hispanic / Latino Asian 185.20 59.50 19.00 S026 20G 55.10 M Non Hispanic / Latino White / Caucasian 161.70 75.30 26.00 S027 22G 29.30 F Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino Asian 155.20 84.20 24.00 S029 20G 44.30 M Non Hispanic / Latino White / Caucasian 170.70 81.60 21.00 S030 20G 52.30 F Non Hispanic / Latino Other 152.50 77.70 25.00 S031 22G 26.50 M Non Hispanic / Latino Asian 178.80 69.60 25.00 S032 22G 45.00 M Non Hispanic / Latino White / Caucasian 166.70 88.70 20.00 S033 22G 28.10 M Non Hispanic / | | | | | | , | 185.30 | | |
| S026 20G 55.10 M Non Hispanic / Latino White / Caucasian 161.70 75.30 26.00 S027 22G 29.30 F Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino Asian 155.20 84.20 24.00 S029 20G 44.30 M Non Hispanic / Latino White / Caucasian 170.70 81.60 21.00 S030 20G 52.30 F Non Hispanic / Latino Other 152.50 77.70 25.00 S031 22G 26.50 M Non Hispanic / Latino Asian 178.80 69.60 25.00 S032 22G 45.00 M Non Hispanic / Latino White / Caucasian 166.70 88.70 20.00 S033 22G 28.10 M Non Hispanic / Latino Other 166.60 63.90 27.00 S034 20G 52.20 F Non Hispanic / | | | | | | | | | |
| S027 22G 29.30 F Non Hispanic / Latino Other 157.00 75.90 19.00 S028 22G 39.10 F Non Hispanic / Latino Asian 155.20 84.20 24.00 S029 20G 44.30 M Non Hispanic / Latino White / Caucasian 170.70 81.60 21.00 S030 20G 52.30 F Non Hispanic / Latino Other 152.50 77.70 25.00 S031 22G 26.50 M Non Hispanic / Latino Asian 178.80 69.60 25.00 S032 22G 45.00 M Non Hispanic / Latino White / Caucasian 166.70 88.70 20.00 S033 22G 28.10 M Non Hispanic / Latino Other 166.60 63.90 27.00 S034 20G 52.20 F Non Hispanic / Latino White / Caucasian 179.50 82.50 21.00 S035 22G 55.50 F Non Hispanic / | S025 | 20G | 28.10 | M | Non Hispanic / Latino | Asian | 185.20 | 59.50 | 19.00 |
| S028 22G 39.10 F Non Hispanic / Latino Asian 155.20 84.20 24.00 S029 20G 44.30 M Non Hispanic / Latino White / Caucasian 170.70 81.60 21.00 S030 20G 52.30 F Non Hispanic / Latino Other 152.50 77.70 25.00 S031 22G 26.50 M Non Hispanic / Latino Asian 178.80 69.60 25.00 S032 22G 45.00 M Non Hispanic / Latino White / Caucasian 166.70 88.70 20.00 S033 22G 28.10 M Non Hispanic / Latino Other 166.60 63.90 27.00 S034 20G 52.20 F Non Hispanic / Latino Asian 169.40 54.70 22.00 S035 22G 55.50 F Non Hispanic / Latino White / Caucasian 179.50 82.50 21.00 S037 20G 55.70 F Non Hispanic / | S026 | 20G | 55.10 | M | Non Hispanic / Latino | White / Caucasian | 161.70 | 75.30 | 26.00 |
| S029 20G 44.30 M Non Hispanic / Latino White / Caucasian 170.70 81.60 21.00 S030 20G 52.30 F Non Hispanic / Latino Other 152.50 77.70 25.00 S031 22G 26.50 M Non Hispanic / Latino Asian 178.80 69.60 25.00 S032 22G 45.00 M Non Hispanic / Latino White / Caucasian 166.70 88.70 20.00 S033 22G 28.10 M Non Hispanic / Latino Other 166.60 63.90 27.00 S034 20G 52.20 F Non Hispanic / Latino Asian 169.40 54.70 22.00 S035 22G 55.50 F Non Hispanic / Latino White / Caucasian 179.50 82.50 21.00 S036 20G 29.90 F Hispanic / Latino Other 153.50 61.10 21.00 S037 20G 55.70 F Non Hispanic / Lat | | | 29.30 | | Non Hispanic / Latino | Other | 157.00 | 75.90 | 19.00 |
| S030 20G 52.30 F Non Hispanic / Latino Other 152.50 77.70 25.00 S031 22G 26.50 M Non Hispanic / Latino Asian 178.80 69.60 25.00 S032 22G 45.00 M Non Hispanic / Latino White / Caucasian 166.70 88.70 20.00 S033 22G 28.10 M Non Hispanic / Latino Other 166.60 63.90 27.00 S034 20G 52.20 F Non Hispanic / Latino Asian 169.40 54.70 22.00 S035 22G 55.50 F Non Hispanic / Latino White / Caucasian 179.50 82.50 21.00 S036 20G 29.90 F Hispanic / Latino Other 153.50 61.10 21.00 S037 20G 55.70 F Non Hispanic / Latino Asian 177.20 73.50 26.00 S038 20G 39.60 M Non Hispanic / Latino | | | 39.10 | F | | Asian | 155.20 | 84.20 | 24.00 |
| S031 22G 26.50 M Non Hispanic / Latino Asian 178.80 69.60 25.00 S032 22G 45.00 M Non Hispanic / Latino White / Caucasian 166.70 88.70 20.00 S033 22G 28.10 M Non Hispanic / Latino Other 166.60 63.90 27.00 S034 20G 52.20 F Non Hispanic / Latino Asian 169.40 54.70 22.00 S035 22G 55.50 F Non Hispanic / Latino White / Caucasian 179.50 82.50 21.00 S036 20G 29.90 F Hispanic / Latino Other 153.50 61.10 21.00 S037 20G 55.70 F Non Hispanic / Latino Asian 177.20 73.50 26.00 S038 20G 39.60 M Non Hispanic / Latino White / Caucasian 154.30 75.80 24.00 S039 22G 23.90 F Non Hispanic / Lat | S029 | 20G | 44.30 | M | Non Hispanic / Latino | White / Caucasian | 170.70 | 81.60 | 21.00 |
| S032 22G 45.00 M Non Hispanic / Latino White / Caucasian 166.70 88.70 20.00 S033 22G 28.10 M Non Hispanic / Latino Other 166.60 63.90 27.00 S034 20G 52.20 F Non Hispanic / Latino Asian 169.40 54.70 22.00 S035 22G 55.50 F Non Hispanic / Latino White / Caucasian 179.50 82.50 21.00 S036 20G 29.90 F Hispanic / Latino Other 153.50 61.10 21.00 S037 20G 55.70 F Non Hispanic / Latino Asian 177.20 73.50 26.00 S038 20G 39.60 M Non Hispanic / Latino White / Caucasian 154.30 75.80 24.00 S039 22G 23.90 F Non Hispanic / Latino Other 158.40 88.60 21.00 | S030 | 20G | 52.30 | F | Non Hispanic / Latino | Other | 152.50 | 77.70 | 25.00 |
| S033 22G 28.10 M Non Hispanic / Latino Other 166.60 63.90 27.00 S034 20G 52.20 F Non Hispanic / Latino Asian 169.40 54.70 22.00 S035 22G 55.50 F Non Hispanic / Latino White / Caucasian 179.50 82.50 21.00 S036 20G 29.90 F Hispanic / Latino Other 153.50 61.10 21.00 S037 20G 55.70 F Non Hispanic / Latino Asian 177.20 73.50 26.00 S038 20G 39.60 M Non Hispanic / Latino White / Caucasian 154.30 75.80 24.00 S039 22G 23.90 F Non Hispanic / Latino Other 158.40 88.60 21.00 | S031 | 22G | 26.50 | M | Non Hispanic / Latino | Asian | 178.80 | 69.60 | 25.00 |
| S034 20G 52.20 F Non Hispanic / Latino Asian 169.40 54.70 22.00 S035 22G 55.50 F Non Hispanic / Latino White / Caucasian 179.50 82.50 21.00 S036 20G 29.90 F Hispanic / Latino Other 153.50 61.10 21.00 S037 20G 55.70 F Non Hispanic / Latino Asian 177.20 73.50 26.00 S038 20G 39.60 M Non Hispanic / Latino White / Caucasian 154.30 75.80 24.00 S039 22G 23.90 F Non Hispanic / Latino Other 158.40 88.60 21.00 | S032 | 22G | 45.00 | M | Non Hispanic / Latino | White / Caucasian | 166.70 | 88.70 | 20.00 |
| S035 22G 55.50 F Non Hispanic / Latino White / Caucasian 179.50 82.50 21.00 S036 20G 29.90 F Hispanic / Latino Other 153.50 61.10 21.00 S037 20G 55.70 F Non Hispanic / Latino Asian 177.20 73.50 26.00 S038 20G 39.60 M Non Hispanic / Latino White / Caucasian 154.30 75.80 24.00 S039 22G 23.90 F Non Hispanic / Latino Other 158.40 88.60 21.00 | S033 | 22G | 28.10 | M | Non Hispanic / Latino | Other | 166.60 | 63.90 | 27.00 |
| S036 20G 29.90 F Hispanic / Latino Other 153.50 61.10 21.00 S037 20G 55.70 F Non Hispanic / Latino Asian 177.20 73.50 26.00 S038 20G 39.60 M Non Hispanic / Latino White / Caucasian 154.30 75.80 24.00 S039 22G 23.90 F Non Hispanic / Latino Other 158.40 88.60 21.00 | S034 | 20G | 52.20 | F | Non Hispanic / Latino | Asian | 169.40 | 54.70 | 22.00 |
| S037 20G 55.70 F Non Hispanic / Latino Asian 177.20 73.50 26.00 S038 20G 39.60 M Non Hispanic / Latino White / Caucasian 154.30 75.80 24.00 S039 22G 23.90 F Non Hispanic / Latino Other 158.40 88.60 21.00 | S035 | 22G | 55.50 | F | Non Hispanic / Latino | White / Caucasian | 179.50 | 82.50 | 21.00 |
| S038 20G 39.60 M Non Hispanic / Latino White / Caucasian 154.30 75.80 24.00 S039 22G 23.90 F Non Hispanic / Latino Other 158.40 88.60 21.00 | S036 | 20G | 29.90 | | Hispanic / Latino | Other | 153.50 | 61.10 | 21.00 |
| S039 22G 23.90 F Non Hispanic / Latino Other 158.40 88.60 21.00 | S037 | 20G | 55.70 | F | Non Hispanic / Latino | Asian | 177.20 | 73.50 | 26.00 |
| 1 / | S038 | 20G | 39.60 | $\mathbf{M}$ | Non Hispanic / Latino | White / Caucasian | 154.30 | 75.80 | 24.00 |
| | S039 | 22G | 23.90 | F | Non Hispanic / Latino | Other | 158.40 | 88.60 | 21.00 |
| 2010 == 2010 11 110 Palito / Davido 110101 10010 00100 20100 | S040 | 22G | 40.90 | $\mathbf{M}$ | Non Hispanic / Latino | Asian | 150.90 | 80.80 | 26.00 |



Table C.0.3: Dummy Family Medical History listing (rows 1 to 40).

| subjID | gauge | bloodDisorderClotting | cancer | heartDisease | highBloodPressure | diabetesType2 |
|---|---|---|---|---|---|---|
| S001 | 22G | No | No | No | No | Yes |
| S002 | 20G | No | No | No | No | No |
| S003 | 20G | No | No | No | No | No |
| S004 | 22G | No | No | No | Yes | No |
| S005 | 22G | Yes | No | No | No | Yes |
| S006 | 20G | No | No | No | Yes | No |
| S007 | 20G | No | No | No | No | No |
| S008 | 22G | Yes | No | No | No | Yes |
| S009 | 22G | No | No | No | No | Yes |
| S010 | 22G | No | No | No | No | No |
| S011 | 20G | No | No | No | No | Yes |
| S012 | 20G | No | No | No | No | No |
| S013 | 20G | No | No | No | Yes | No |
| S014 | 22G | No | No | No | No | No |
| S015 | 20G | No | No | No | Yes | No |
| S016 | 22G | No | No | No | No | No |
| S017 | 20G | No | No | No | Yes | No |
| S018 | 22G | No | No | No | No | No |
| S019 | 22G | No | No | No | No | No |
| S020 | 20G | No | No | No | Yes | No |
| S021 | 22G | No | No | No | No | No |
| S022 | 20G | No | Yes | No | Yes | No |
| S023 | 22G | No | No | No | No | No |
| S024 | 20G | No | No | No | No | No |
| S025 | 20G | No | No | No | Yes | No |
| S026 | 20G | No | No | No | No | No |
| S027 | 22G | No | No | No | No | Yes |
| S028 | 22G | No | Yes | No | No | No |
| S029 | 20G | No | No | No | No | No |
| S030 | 20G | No | No | No | No | No |
| S031 | 22G | No | No | No | No | No |
| S032 | 22G | No | No | No | No | No |
| S033 | 22G | No | No | No | No | No |
| S034 | 20G | No | No | No | No | No |
| S035 | 22G | No | No | No | No | Yes |
| S036 | 20G | No | No | No | No | No |
| S037 | 20G | No | No | No | No | No |
| S038 | 20G | No | No | No | No | No |
| S039 | 22G | No | No | No | No | No |
| S040 | 22G | No | No | No | No | No |



Table C.0.4: Dummy Baseline listing (rows 1 to 40).

| | 0.0.4. | Dunning Das | - \ | JWS I IC | , 40). |
|--------|--------|--------------|----------------|----------|-------------|
| subjID | gauge | tipMidStream | tipWallContact | bfv | $cv\_ratio$ |
| S001 | 22G | Yes | No | 162.86 | 35.70 |
| S002 | 20G | Yes | No | 169.78 | 33.96 |
| S003 | 20G | Yes | Yes | 157.73 | 39.69 |
| S004 | 22G | Yes | Yes | 151.31 | 42.67 |
| S005 | 22G | No | No | 165.24 | 36.42 |
| S006 | 20G | No | No | 164.16 | 44.91 |
| S007 | 20G | Yes | No | 168.51 | 35.11 |
| S008 | 22G | No | No | 163.64 | 30.23 |
| S009 | 22G | Yes | No | 173.14 | 33.27 |
| S010 | 22G | Yes | No | 164.40 | 40.57 |
| S011 | 20G | Yes | No | 159.85 | 41.06 |
| S012 | 20G | No | No | 173.71 | 37.45 |
| S013 | 20G | Yes | Yes | 160.25 | 42.14 |
| S014 | 22G | Yes | No | 166.91 | 31.00 |
| S015 | 20G | Yes | No | 155.56 | 44.65 |
| S016 | 22G | Yes | No | 159.83 | 35.38 |
| S017 | 20G | Yes | No | 163.14 | 42.58 |
| S018 | 22G | Yes | No | 161.69 | 38.99 |
| S019 | 22G | No | No | 159.15 | 34.75 |
| S020 | 20G | Yes | No | 151.37 | 43.20 |
| S021 | 22G | Yes | No | 163.94 | 34.72 |
| S022 | 20G | Yes | Yes | 169.70 | 42.95 |
| S023 | 22G | No | No | 164.49 | 40.26 |
| S024 | 20G | Yes | No | 161.92 | 32.11 |
| S025 | 20G | Yes | No | 173.03 | 42.02 |
| S026 | 20G | No | No | 154.34 | 33.76 |
| S027 | 22G | Yes | Yes | 155.45 | 41.91 |
| S028 | 22G | Yes | Yes | 155.20 | 30.45 |
| S029 | 20G | Yes | No | 169.53 | 33.37 |
| S030 | 20G | Yes | No | 157.41 | 35.70 |
| S031 | 22G | Yes | No | 150.97 | 33.86 |
| S032 | 22G | Yes | No | 157.20 | 33.50 |
| S033 | 22G | Yes | No | 158.89 | 33.09 |
| S034 | 20G | Yes | Yes | 161.70 | 38.45 |
| S035 | 22G | No | No | 173.17 | 39.35 |
| S036 | 20G | Yes | No | 158.18 | 39.31 |
| S037 | 20G | No | No | 150.46 | 33.90 |
| S038 | 20G | Yes | No | 158.48 | 37.64 |
| S039 | 22G | Yes | No | 173.28 | 40.17 |
| S040 | 22G | Yes | No | 156.54 | 32.07 |



Table C.0.5: Dummy Indwell Time listing (rows 1 to 40).

| subjID | device | lifeTime | indwellTime_cont | status | eventType | indwellTime_disc |
|---|---|---|---|---|---|---|
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 1.00 | blood_draw_6mL | 72.00 |
| S001 | BD Nexiva (22G x 1 inch) BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 1.00 | blood_draw_6mL | 72.00 |
| S002 | BD Nexiva (20G x 1 inch) | 80.58 | 72.00 | 0.00 | biood_draw_com2 | 72.00 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 1.00 | flush | 72.00 |
| S003 | BD Nexiva (20G x 1 inch) | 57.79 | 57.79 | 1.00 | blood_draw_6mL | 54.00 |
| S003 | BD Nexiva (20G x 1.75 inch) | 91.75 | 72.00 | 0.00 | biood_draw_omiL | 72.00 |
| S004 | BD Nexiva (22G x 1 inch) | 66.26 | 66.26 | 0.00 | | 72.00 |
| S004 | BD Nexiva (22G x 1.75 inch) | 86.02 | 72.00 | 1.00 | flush | 72.00 |
| S005 | BD Nexiva (22G x 1 inch) | 90.85 | 72.00 | 0.00 | | 72.00 |
| S005 | BD Nexiva (22G x 1.75 inch) | 66.75 | 66.75 | 1.00 | flush | 72.00 |
| S006 | BD Nexiva (20G x 1 inch) | 64.59 | 64.59 | 0.00 | | 72.00 |
| S006 | BD Nexiva (20G x 1.75 inch) | 69.34 | 69.34 | 0.00 | | 72.00 |
| S007 | BD Nexiva (20G x 1 inch) | 61.96 | 61.96 | 1.00 | flush | 54.00 |
| S007 | BD Nexiva (20G x 1.75 inch) | 72.67 | 72.00 | 0.00 | | 72.00 |
| S008 | BD Nexiva (22G x 1 inch) | 35.96 | 35.96 | 1.00 | flush | 30.00 |
| S008 | BD Nexiva (22G x 1.75 inch) | 95.55 | 72.00 | 0.00 | | 72.00 |
| S009 | BD Nexiva (22G x 1 inch) | 37.24 | 37.24 | 1.00 | $blood\_draw\_2mL$ | 30.00 |
| S009 | BD Nexiva (22G x 1.75 inch) | 22.31 | 22.31 | 1.00 | $blood\_draw\_2mL$ | 24.00 |
| S010 | BD Nexiva (22G x 1 inch) | 28.76 | 28.76 | 0.00 | | 30.00 |
| S010 | BD Nexiva (22G x 1.75 inch) | 44.98 | 44.98 | 1.00 | flush | 48.00 |
| S011 | BD Nexiva (20G x 1 inch) | 43.29 | 43.29 | 1.00 | flush | 48.00 |
| S011 | BD Nexiva (20G x 1.75 inch) | 93.55 | 72.00 | 0.00 | | 72.00 |
| S012 | BD Nexiva (20G x 1 inch) | 37.93 | 37.93 | 0.00 | | 30.00 |
| S012 | BD Nexiva (20G x 1.75 inch) | 83.98 | 72.00 | 0.00 | | 72.00 |
| S013 | BD Nexiva (20G x 1 inch) | 74.79 | 72.00 | 1.00 | flush | 72.00 |
| S013 | BD Nexiva (20G x 1.75 inch) | 70.04 | 70.04 | 0.00 | | 72.00 |
| S014 | BD Nexiva (22G x 1 inch) | 73.05 | 72.00 | 1.00 | $blood\_draw\_2mL$ | 72.00 |
| S014 | BD Nexiva (22G x 1.75 inch) | 70.67 | 70.67 | 0.00 | | 72.00 |
| S015 | BD Nexiva (20G x 1 inch) | 53.34 | 53.34 | 1.00 | $blood\_draw\_2mL$ | 54.00 |
| S015 | BD Nexiva (20G x 1.75 inch) | 92.07 | 72.00 | 1.00 | flush | 72.00 |
| S016 | BD Nexiva (22G x 1 inch) | 10.73 | 10.73 | 1.00 | flush | 6.00 |
| S016 | BD Nexiva (22G x 1.75 inch) | 61.41 | 61.41 | 0.00 | | 54.00 |
| S017 | BD Nexiva (20G x 1 inch) | 68.60 | 68.60 | 0.00 | | 72.00 |
| S017 | BD Nexiva (20G x 1.75 inch) | 58.60 | 58.60 | 1.00 | flush | 54.00 |
| S018 | BD Nexiva (22G x 1 inch) | 43.54 | 43.54 | 1.00 | $blood\_draw\_6mL$ | 48.00 |
| S018 | BD Nexiva (22G x 1.75 inch) | 64.02 | 64.02 | 1.00 | flush | 72.00 |
| S019 | BD Nexiva (22G x 1 inch) | 26.92 | 26.92 | 1.00 | flush | 24.00 |
| S019 | BD Nexiva (22G x 1.75 inch) | 82.65 | 72.00 | 0.00 | | 72.00 |
| S020 | BD Nexiva (20G x 1 inch) | 73.47 | 72.00 | 1.00 | $blood\_draw\_2mL$ | 72.00 |
| S020 | BD Nexiva (20G x 1.75 inch) | 87.35 | 72.00 | 0.00 | | 72.00 |

Table C.0.6: Dummy Blood Analysis listing (rows 1 to 40).

| | Table C.0.6: Dummy Blood Analysis listing (rows 1 to 40). | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| subjID | device | lifeTime | Indwell | Indwell | baselineCfHb | timepoint | tube | cfHb | haemolysis | haemolysis | Blood |
| | | | Time | Time | | | | | - AU480 | - Visual | Draw |
| | | | (cont.) | (cat.) | | | | | | | Duration |
| | | | | | | | | | | | (sec.) |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 0.00 | 2mL | 143.26 | No | No | 62.52 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 0.00 | 6mL | 189.17 | No | Yes | 102.54 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 6.00 | 2mL | 149.51 | No | No | 59.28 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 6.00 | 6mL | 198.38 | No | Yes | 84.14 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 24.00 | 2mL | 198.79 | No | Yes | 62.80 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 24.00 | 6mL | 146.22 | No | No | 102.12 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 30.00 | 2mL | 216.39 | Yes | Yes | 59.31 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 30.00 | 6mL | 191.83 | No | Yes | 105.70 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 48.00 | 2mL | 215.34 | Yes | Yes | 59.57 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 48.00 | 6mL | 284.53 | Yes | Yes | 94.84 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 54.00 | 2mL | 162.19 | No | No | 65.32 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 54.00 | 6mL | 169.64 | No | No | 103.54 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 72.00 | 2mL | 152.62 | No | No | 64.50 |
| S001 | BD Nexiva (22G x 1 inch) | 67.20 | 67.20 | 72.00 | 191.86 | 72.00 | 6mL | 156.91 | No | No | 94.85 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 0.00 | 2mL | 153.01 | No | No | 57.46 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 0.00 | 6mL | 186.75 | No | Yes | 109.77 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 6.00 | 2mL | 168.11 | No | No | 56.58 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 6.00 | 6mL | 161.64 | No | No | 109.21 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 24.00 | 2mL | 195.47 | No | Yes | 53.42 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 24.00 | 6mL | 163.25 | No | No | 107.81 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 30.00 | 2mL | 202.26 | Yes | Yes | 59.02 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 30.00 | 6mL | 171.86 | No | No | 101.98 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 48.00 | 2mL | 135.55 | No | No | 61.49 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 48.00 | 6mL | 174.44 | No | No | 97.01 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 54.00 | 2mL | 114.32 | No | No | 49.53 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 54.00 | 6mL | 163.32 | No | No | 106.43 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 72.00 | 2mL | 217.83 | Yes | Yes | 64.70 |
| S001 | BD Nexiva (22G x 1.75 inch) | 72.53 | 72.00 | 72.00 | 191.86 | 72.00 | 6mL | 148.19 | No | No | 105.51 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 0.00 | 2mL | 153.96 | No | No | 54.68 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 0.00 | 6mL | 153.11 | No | No | 95.97 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 6.00 | 2mL | 153.49 | No | No | 64.35 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 6.00 | 6mL | 205.98 | Yes | Yes | 96.23 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 24.00 | 2mL | 130.04 | No | No | 62.57 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 24.00 | 6mL | 161.20 | No | No | 104.41 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 30.00 | 2mL | 139.05 | No | No | 68.95 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 30.00 | 6mL | 158.97 | No | No | 95.09 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 48.00 | 2mL | 155.15 | No | No | 59.26 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 48.00 | 6mL | 140.26 | No | No | 95.75 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 54.00 | 2mL | 160.11 | No | No | 61.84 |
| S002 | BD Nexiva (20G x 1.75 inch) | 68.25 | 68.25 | 72.00 | 176.53 | 54.00 | $6 \mathrm{mL}$ | 149.46 | No | No | 94.52 |





Table C.0.7: Dummy Blood Analysis Baseline listing (rows 1 to 40).

| subjID | gauge | tube | cfHb | haemolysis_AU480 | haemolysis_Visual | bloodDrawDuration |
|---|---|---|---|---|---|---|
| S001 | 22G | 2mL | 148.74 | No | No | 43.72 |
| S001 | 22G | $6 \mathrm{mL}$ | 234.99 | Yes | Yes | 111.18 |
| S002 | 20G | 2mL | 224.05 | Yes | Yes | 32.77 |
| S002 | 20G | 6 mL | 129.02 | No | No | 104.25 |
| S003 | 20G | 2mL | 212.55 | Yes | Yes | 33.82 |
| S003 | 20G | $6 \mathrm{mL}$ | 263.10 | Yes | Yes | 86.61 |
| S004 | 22G | 2mL | 135.19 | No | No | 40.63 |
| S004 | 22G | $6 \mathrm{mL}$ | 259.57 | Yes | Yes | 98.93 |
| S005 | 22G | 2mL | 202.30 | Yes | Yes | 37.65 |
| S005 | 22G | $6 \mathrm{mL}$ | 244.32 | Yes | Yes | 100.27 |
| S006 | 20G | 2mL | 223.75 | Yes | Yes | 42.84 |
| S006 | 20G | $6 \mathrm{mL}$ | 216.52 | Yes | Yes | 95.40 |
| S007 | 20G | 2mL | 56.99 | No | No | 43.10 |
| S007 | 20G | $6 \mathrm{mL}$ | 225.63 | Yes | Yes | 102.07 |
| S008 | 22G | 2mL | 148.56 | No | No | 35.68 |
| S008 | 22G | $6 \mathrm{mL}$ | 185.07 | No | Yes | 100.02 |
| S009 | 22G | 2mL | 197.34 | No | Yes | 42.94 |
| S009 | 22G | $6 \mathrm{mL}$ | 311.35 | Yes | Yes | 92.57 |
| S010 | 22G | 2mL | 210.10 | Yes | Yes | 42.49 |
| S010 | 22G | 6 mL | 262.42 | Yes | Yes | 97.18 |
| S011 | 20G | 2mL | 197.32 | No | Yes | 42.06 |
| S011 | 20G | 6 mL | 143.21 | No | No | 93.79 |
| S012 | 20G | 2mL | 264.69 | Yes | Yes | 36.38 |
| S012 | 20G | 6 mL | 210.89 | Yes | Yes | 88.81 |
| S013 | 20G | 2mL | 196.52 | No | Yes | 36.05 |
| S013 | 20G | 6 mL | 219.72 | Yes | Yes | 104.09 |
| S014 | 22G | 2mL | 124.86 | No | No | 43.14 |
| S014 | 22G | 6 mL | 197.42 | No | Yes | 106.31 |
| S015 | 20G | 2mL | 132.21 | No | No | 42.66 |
| S015 | 20G | 6 mL | 214.86 | Yes | Yes | 108.96 |
| S016 | 22G | 2mL | 237.06 | Yes | Yes | 38.79 |
| S016 | 22G | $6 \mathrm{mL}$ | 167.25 | No | No | 101.38 |
| S017 | 20G | 2mL | 191.75 | No | Yes | 42.19 |
| S017 | 20G | 6 mL | 275.98 | Yes | Yes | 103.73 |
| S018 | 22G | 2mL | 171.68 | No | No | 32.80 |
| S018 | 22G | 6 mL | 227.78 | Yes | Yes | 91.10 |
| S019 | 22G | 2mL | 155.16 | No | No | 44.12 |
| S019 | 22G | $6 \mathrm{mL}$ | 165.42 | No | No | 116.40 |
| S020 | 20G | 2mL | 204.74 | Yes | Yes | 41.08 |
| S020 | 20G | $6 \mathrm{mL}$ | 216.52 | Yes | Yes | 94.47 |





#### $\mathbf{D}$ **Additional Figures**

#### D.1 **PIVC Rescue Decision Tree**

**FLUSH PROCEDURES** Attachment 1: Decision Tree Flowchart CAN CATHETER BE FLUSHED? Conduct observation for infiltration at each flush attempt IS THERE ANY LEAKAGE? **ENSURE LUER CONNECTION** ARE THE CLAMPS LOCKED?
IS EXTENSION SET KINKED/IMPINGED? CAN CATHETER BE FLUSHED? RELEASE CLAMPS ATTEMPT TO UNKINK EXTENSION SET VISUAL SIGN OF CATHETER DISLODGEMENT THROUGH DRESSING? CAN CATHETER BE FLUSHED? VISUAL SIGN OF CATHETER KINK THROUGH THE DRESSING REMOVE DRESSING, APPLY NEW DRESSING CAN CATHETER BE FLUSHED? HEATPACK TO FOREARM/HAND FOR ~5 MIN CAN CATHETER BE FLUSHED? VASOSPASM/THROMBUS OBSERVED VIA COLOR DUPLEX ULTRASOUND? REMOVE PIVC Evaluate for Device Deficiency

Figure D.1.1: PIVC Rescue Decision Tree for Flush Procedures





Figure D.1.2: PIVC Rescue Decision Tree for Aspiration Procedures